

Title: An Open-Label, Extension Study of Teduglutide in Japanese Subjects with Short Bowel Syndrome who Completed 24 Weeks of Treatment in SHP633-306 or TED-C14-004

NCT Number: NCT03596164

Protocol Approve Date: 06-Nov-2020

Certain information within this protocol has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).



PROTOCOL: SHP633-307

ble Letins of Use An Open-Label, Extension Study of Teduglutide in Japanese Subjects TITLE:

of I all subject to the all with Short Bowel Syndrome who Completed 24 Weeks of Treatment in

SHP633-306 or TED-C14-004

SHP633-307 **NUMBER** 

**PHASE** 3 Extension

**DRUG:** Teduglutide

Short bowel syndrome **INDICATION:** 

Shire Human Genetic Therapies, Inc. **SPONSOR:** 

Takeda Pharmaceutical Company Limited

1-1, Doshomachi 4-Chrome, Chuo-ku, Osaka-shi

Osaka Japan

Amendment 2: 06 Nov 2020 **PROTOCOL** 

Origina Origina Property of Takedai. For non-co **HISTORY:** Amendment 1: 27 Sep 2018

Original Protocol: 23 Jan 2018

## PROTOCOL SIGNATURE PAGE

| <b>Date:</b> 10-Nov-2020 12:28 EST |
|--------------------------------------|
| ∠e <sup>s</sup> |

## Investigator's Acknowledgement

I have read this protocol for Shire Study SHP633-307.

**Title:** An Open-Label, Extension Study of Teduglutide in Japanese Subjects with Short Bowel Syndrome who Completed 24 Weeks of Treatment in SHP633-306 or TED ©14-004

I have fully discussed the objective(s) of this study and the contents of this protocol with the sponsor's representative.

I understand that the information in this protocol is confidential and should not be disclosed, other than to those directly involved in the execution or the scientific/ethical review of the study, without written authorization from the sponsor. It is, however, permissible to provide the information contained herein to a subject in order to obtain their consent to participate.

I agree to conduct this study according to this protocol and to comply with its requirements, subject to ethical and safety considerations and guidelines, and to conduct the study in accordance with International Conference on Harmonization (ICH) guidelines on Good Clinical Practice (GCP) and with the applicable regulatory requirements.

I understand that failure to comply with the requirements of the protocol may lead to the termination of my participation as an investigator for this study.

I understand that the sponsor may decide to suspend or prematurely terminate the study at any time for whatever reason; such a decision will be communicated to me in writing. Conversely, should I decide to withdraw from execution of the study I will communicate my intention immediately in writing to the sponsor.

| Investigator Name and<br>Address: | |
|-----------------------------------|-------|
| (please hand print or type) | |
| Signature: | Date: |

# SUMMARY OF CHANGES FROM PREVIOUS PROTOCOL VERSION

| Protocol Amendments | | |
|---|---|---|
| Summary of Change(s) Since the Last Version of the Approved Protocol | | |
| Amendment Number 2 | Amendment Date<br>06 Nov 2020 | Global |
| Description of Change and Rationa | le | Section(s) Affected by Change |
| Sponsor Name Changed to include both Shire Human Genetic Therapies, Inc. (USA) and Takeda Pharmaceutical Company Limited The Sponsor name was updated to align more accurately with legal entities responsible for study. | | Signature Page |
| Changed name of sponsor protocol si | gnatory to | Signature Page |
| Transferred back the role of in-country Services Japan K.K to the sponsor. To notifying the relevant regulatory authoracy adverse events. | Emergency Contact Information<br>Section 8.2.7 | |
| Changed the name of the Shire medic | al monitor to | Emergency Contact Information |
| Updated the Shire medical monitor conumbers; the fax number was remove Clarified the timeframe for calling the to 20:00 US Eastern Standard Time. (Administrative Amendments dated 1) | | |
| Specified that the SHP633-307 study study if teduglutide is approved for m | Section 3.2 | |
| Clarified that the short term prescript 72 hours should be recorded in the clamedications, not as PN/IV adjustmen (Administrative Amendment dated) | Section 5.1 | |
| Added a new section entitled "Chang | es to Study Procedures Due to a<br>nges is to maintain the subject safety,<br>the context of healthcare delivery | Section 7.3 |
| Clarified the definition of an overdos investigational product at a dose or fr subcutaneous once daily. An overdos criteria are met: • More than 0.05 mg/kg is given a: • Consecutive doses are spaced les • Any more than 0.05 mg/kg in on 12:00 AM and ending at 11:59 PM (Clarification Memo dated 12 Jun 20 | equency greater than 0.05 mg/kg e occurs if any of the following t any one time as than 12 hours apart e day (a day is defined as beginning at f) | Section 8.1.7 |
| Clarified that the next scheduled visit not from Visit 1. | should be based on the previous visit, | Table 1 (a note was added) Table 2 (a note was added) |
| (Clarification Memo dated 18 Dec 20 | 119) | Section 7.1 |

| | Protocol Amendments | |
|---|---|---|
| | hange(s) Since the Last Version of the | |
| Amendment Number<br>2 | Amendment Date<br>06 Nov 2020 | Global |
| Description of Change and Ration | nale | Section(s) Affected by Chang |
| 48-hour Urinary Output (scheduled parenteral nutrition action to be take 1.0 L/day or the target based on stal | | iical) <sup>k</sup> |
| Corrections to typographical errors intent of the original document) were | (which do not modify content and/or | Throughout the protocol |
| of non-cox | (which do not modify content and/or re made. | |
| of Takedai. For non-cor | | |

## EMERGENCY CONTACT INFORMATION

In the event of a serious adverse event (SAE), the investigator must fax or e-mail the Shire Clinical Study Adverse Event Form for Serious Adverse Events and Non-serious AEs as Required by Protocol within 24 hours to the sponsor or designee using the details below. Applicable fax numbers and e-mail address can also be found on the form (sent under separate cover).



## PRODUCT QUALITY COMPLAINTS

einsoiuse Investigators are required to report investigational product quality complaints to Shire within 24 hours. This includes any instances wherein the quality or performance of a Shire product (marketed or investigational) does not meet expectations (eg, inadequate or faulty closure, product contamination) or that the product did not meet the specifications defined in the application for the product (eg, wrong product such that the label and contents are different products). For instructions on reporting AEs related to product complaints, see Section 8.

The product quality includes quality of the drug delivery device combination product. As such device defects should be reported according to the instructions in this section. The reporting of product quality occurrences, when the product does not meet specifications, includes the reporting of device defects.

Please use the information below as applicable to report the Product Quality Complaint:

| Origin of Product Quality Complaint | E-mail Address |
|-------------------------------------|----------------|
| | · |
| European Union and Rest of World | |
| | . 5 |

ce, if nee of a room, commercial use of a ro Telephone numbers (provided for reference, if needed):

# TABLE OF CONTENTS

| PROTOCOL SIGNATURE PAGE | 2 |
|---|---|
| SUMMARY OF CHANGES FROM PREVIOUS PROTOCOL VERSION | |
| EMERGENCY CONTACT INFORMATION | |
| PRODUCT QUALITY COMPLAINTS | / |
| TABLE OF CONTENTS | 4 (2) |
| LIST OF TABLES | |
| LIST OF FIGURES | 11 |
| LIST OF APPENDICES | 11 |
| LIST OF FIGURESLIST OF APPENDICESLIST OF ABBREVIATIONS AND DEFINITION OF TERMS | |
| STUDY SYNOPSIS | <b>©</b> 13 |
| STUDY SCHEDULES | 16 |
| STUDY SCHEDULES | 21 |
| 1.1 Indication and Current Treatment Options | 21 |
| 1.2 Product Background and Clinical Information | 22 |
| 2 STUDY OBJECTIVES AND PURPOSE 2.1 Rationale for the Study | 24 |
| 2.1 Rationale for the Study | 24 |
| 2.2 Study Objectives | 24 |
| 2.2 Study Objectives | 25 |
| 3.1 Study Design and Flow Chart | 25 |
| 3.2 Duration and Study Completion Definition | 25 |
| 3.3 Sites and Regions C | 25 |
| 4 STUDY POPULATION | 27 |
| 4.1 Inclusion Cateria | 27 |
| 4.2 Exclusion Criteria | 27 |
| 4.3 Reproductive Potential | 27 |
| 4.4 Discontinuation of Subjects | 27 |
| 4.4.1 Reasons for Discontinuation | 28 |
| 4.4.2 Subjects "Lost to Follow-up" Prior to Last Scheduled Visit | 28 |
| 5 CONCOMITANT TREATMENT | 29 |
| Concomitant Treatment | 29 |
| 5.1.1 Permitted Treatment | 29 |
| 5.1.2 Prohibited Treatment | 29 |
| 6 INVESTIGATIONAL PRODUCT | 30 |
| 6.1 Identity of Investigational Product | 30 |
| 6.1.1 Blinding the Treatment Assignment | 30 |
| 6.2 Administration of Investigational Product | 30 |

| Silire |
|---------------------------------|
| SHP633-307 Protocol Amendment 2 |
| Teduglutide |

| occ 507 I Totocoi / Imenament 2 | |
|---------------------------------|-------------|
| uglutide | 06 Nov 2020 |

| | 8 | | |
|---|---|---|---|
| | 6.2.1 | Allocation of Subjects to Treatment | 30 |
| | 6.2.2 | Dosing | 30 |
| | 6.2 | 2.2.1 Subject Administration | 30 |
| | 6.2.3 | Unblinding the Treatment Assignment | 31 |
| | 6.3 | Labeling, Packaging, Storage, and Handling | 31 |
| | 6.3.1 | Labeling and Packaging | \$1 |
| | 6.3.2 | Storage and Handling | 32 |
| | 6.4 | Storage and Handling Drug Accountability Subject Compliance PROCEDURES Study Schedule First Visit Treatment Period | 33 |
| | 6.5 | Subject Compliance | 34 |
| 7 | STUDY | PROCEDURES | 35 |
| | 7.1 | Study Schedule | 35 |
| | 7.1.1 | First Visit | 35 |
| | 7.1.2 | Treatment Period. | 35 |
| | 7.2 | Study Evaluations and Procedures | 35 |
| | 7.2.1 | Efficacy Assessments | 35 |
| | 7.2 | Study Evaluations and Procedures Efficacy Assessments 2.1.1 Subject Diaries 2.1.2 Prescribed Parenteral Nutrition | 35 |
| | 7.2 | 2.1.2 Prescribed Parenteral Nutrition | 36 |
| | 7.2 | 2.1.3 Plasma Citrulline | 36 |
| | 7.2.2 | 2.1.2 Prescribed Parenteral Nutrition 2.1.3 Plasma Citrulline Safety Assessments 2.2.1 Laboratory Evaluations | 36 |
| | 7.2 | 2.2.1 Laboratory Evaluations | 36 |
| | 7.2 | 2.2.2 Antibodies to Teduglutide | 37 |
| | 7.2 | 2.2.3 Physical Examinations | 38 |
| | 7.2 | 2.2.4 Vital Signs, Body Weight, and Height | 38 |
| | 7.2 | 2.2.5 Electrocardiograms | |
| | 7.2 | 2.2.6 Gastrointestinal-specific Testing | 38 |
| | 7.2 | 2.2.7 48-Hour Oral Fluid Intake and Urine Output | |
| | 7.2.3 | Pharmacokinetic Assessments | 39 |
| | 7.3 | Changes to Study Procedures Due to a Pandemic | 40 |
| 8 | ADVER\$ | SE AND SERIOUS ADVERSE EVENTS ASSESSMENT | |
| | 8.1 | Definition of Adverse Events, Period of Observation, Recording of | |
| | W. C. | Adverse Events | |
| C | 8.1.1 | Severity Categorization | |
| Ó | 8.1.2 | Relationship Categorization | |
| | 8.1.3 | Outcome Categorization | |
| | 8.1.4 | Symptoms of the Disease under Study | |
| | 8.1.5 | Clinical Laboratory and Other Safety Evaluations | |
| | 8.1.6 | Pregnancy | |
| | 8.1.7 | Abuse, Misuse, Overdose, and Medication Error | 45 |

| Sinc |
|---------------------------------|
| SHP633-307 Protocol Amendment 2 |
| Teduglutide |

| 06 | Nov | 1 | ഹ | n |
|----|------|---|-----|---|
| vv | INUV | 4 | UZ. | U |

| | 8.2 | Serious Adverse Event Procedures | 46 |
|---|---|---|---|
| | 8.2.1 | Reference Safety Information | 46 |
| | 8.2.2 | Reporting Procedures | 46 |
| | 8.2.3 | Serious Adverse Event Definition | 46 |
| | 8.2.4 | Serious Adverse Event Collection Time Frame | 47 |
| | 8.2.5 | Serious Adverse Event Onset and Resolution Dates | 47 |
| | 8.2.6 | Fatal Outcome | 47 |
| | 8.2.7 | Regulatory Agency, Institutional Review Board, Ethics Committee, and Site | 47 |
| | 8.3 | Reporting | 48 |
| 9 | DATA N | MANAGEMENT AND STATISTICAL METHODS | 49 |
| | 9.1 | Data Collection | 49 |
| | 9.2 | Clinical Data Management Statistical Analysis Process Planned Interim Analysis Sample Size Calculation and Power Considerations | 49 |
| | 9.3 | Statistical Analysis Process | 49 |
| | 9.4 | Planned Interim Analysis | 49 |
| | 9.5 | Sample Size Calculation and Power Considerations | 50 |
| | 9.6 | Study Population | 50 |
| | 9.7 | Efficacy Analyses | 50 |
| | 9.8 | Safety Analyses | 51 |
| | 9.9 | Study Population Efficacy Analyses Safety Analyses Pharmacokinetics Analyses | 51 |
| 10 | | OR'S AND INVESTIGATOR'S RESPONSIBILITIES | 52 |
| | 10.1 | Sponsor's Responsibilities | |
| | 10.1. | 1 Good Clinical Practice Compliance | |
| | | 2 Indemnity/Liability and Insurance | |
| | | Public Posting of Study Information | |
| | | 4 Submission of Summary of Clinical Study Report to Competent Authorities | |
| | 10.1 | of Member States Concerned and Ethics Committees | |
| | 10.1 | Investigator's Responsibilities | |
| | | Good Clinical Practice Compliance | |
| | | 2 Protocol Adherence and Investigator Agreement | |
| | V- | 3 Documentation and Retention of Records | |
| ٤ | | 0.2.3.1 Electronic Case Report Forms | |
| O, | | 0.2.3.2 Recording, Access, and Retention of Source Data and Study | |
| | 10 | Documents | 54 |
| | 10 | 0.2.3.3 Audit/Inspection | |
| | 10 | 0.2.3.4 Financial Disclosure | |
| | 10.3 | Ethical Considerations | 55 |

# LIST OF TABLES

| Table 1 | Schedule of Evaluations and Procedures for Subjects Enrolling from SHP633-306 |
|---|---|
| Table 2 | Schedule of Evaluations and Procedures – For Subjects Enrolling from TED-C14-004 |
| Table 3 | TED-C14-004 19 Prohibited Treatment 29 |
| Table 4 | List of Laboratory Tests |
| | LIST OF FIGURES SHP633-307 Study Schematic 26 |
| Figure 1 | SHP633-307 Study Schematic |
| Appendix 1 | |
| Appendix 2 | |
| Property of Takeda. F | or non-commercial use only all |

# LIST OF ABBREVIATIONS AND DEFINITION OF TERMS

| | Abbreviation | Definition |
|---|---|---|
| | AE | adverse event |
| | AUC | area under the plasma concentration-time curve |
| | $AUC_{0-t}$ | AUC from zero to the last measurable concentration |
| | BUN | blood urea nitrogen |
| | CL/F | apparent clearance |
| | $C_{\text{max}}$ | maximum plasma concentration |
| | COVID-19 | coronavirus disease 2019 |
| | CRO | contract research organization |
| | ECG | electrocardiogram |
| | eCRF | electronic case report form |
| | EGD | esophagogastroduodenoscopy |
| | EMA | European Medicines Agency |
| | EOT | end of treatment |
| | EU | European Union |
| | FDA | Food and Drug Administration |
| | GCP | Good Clinical Practice |
| | GI | apparent clearance maximum plasma concentration coronavirus disease 2019 contract research organization electrocardiogram electronic case report form esophagogastroduodenoscopy European Medicines Agency end of treatment European Union Food and Drug Administration Good Clinical Practice gastrointestinal glucagon-like peptide International Committee of Medicinal Journal Editors |
| | GLP | glucagon-like peptide |
| | ICMJE | International Committee of Medicinal Journal Editors |
| | ICH | International Committee on Harmonisation |
| | I/O | oral fluid intake and urine output |
| | IRB | Institutional Review Board |
| | IV | intravenous |
| | MedDRA | Medical Dictionary for Regulatory Activities |
| | PK | pharmacokinetics |
| | PN/IV | parenteral nutrition/intraveneous |
| | PNALD | parenteral nutrition-associated liver disease |
| | SAE | serious adverse event |
| | SAP | statistical analysis plan |
| | SAE SAP SBS SC | short bowel syndrome |
| | SC | subcutaneous |
| | <b>t</b> <sub>1/2</sub> | terminal-phase half-life |
| ( | $t_{\rm max}$ | time to C <sub>max</sub> |
| ) | ULN | upper limit of normal |
| | US | United States |
| | V/F | apparent volume of distribution |

#### STUDY SYNOPSIS

**Protocol number:** SHP633-307 **Drug:** Teduglutide

**Title of the study:** An Open-Label, Extension Study of Teduglutide in Japanese Subjects with Short Bowel Syndrome who Completed 24 Weeks of Treatment in SHP633-306 or TED-C14-004

#### Number of subjects (total and for each treatment arm):

Approximately 5 subjects who completed Study SHP633-306 and up to 7 subjects in TED-C14-004 may enroll in this extension study.

**Investigator(s):** Multicenter study.

#### Site(s) and Region(s):

This study is planned to be conducted in approximately 5 sites in Japan.

| Study period (planned): | Clinical phase: | 3 Extension |
|-------------------------|-----------------|-------------|
| 2018-2021 | | Ċ, |

#### **Objectives:**

The objectives of this clinical study are to evaluate the long-term safety and efficacy of teduglutide in Japanese subjects with parenteral nutrition/intravenous (PN/IV)-dependent short bowel syndrome (SBS) who completed SHP633-306 or who were in the extension phase of TED-C14-004 study.

#### Investigational product, dose, and mode of administration:

Teduglutide 0.05 mg/kg subcutaneously (SC) once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm.

The Site Training Guide specifies the process for training subjects and measures to be taken to provide oversight on study drug administration.

#### Methodology:

This will be a long-term extension study to evaluate the safety and efficacy of teduglutide in Japanese subjects who completed Study SHP633-306 or were in the extension phase of TED-C14-004 (core studies).

Once informed consent has been obtained, demographics, updates to medical history and short bowel syndrome history will be obtained. Teduglutide 0.05 mg/kg will be administered once daily until teduglutide is commercially available, or the subject's participation in this study is discontinued, or the study is discontinued. At each site visit, efficacy (adjustments to PN/IV) and safety will be monitored.

For subjects transitioning from SHP633-306, the SHP633-306 EOS visit assessments will be combined with the assessments for the first visit in SHP633-307. Clinic and phone visits will then alternate on a monthly basis through Month 24; thereafter, clinic visits will occur every 3 months. For subjects transitioning from TED-C14-004, the TED-C14-004 EOS visit assessments will be combined with the assessments for the first visit in SHP633-307; thereafter clinic visits will occur every 3 months.

Subjects enrolling from TED-C14-004 will have blood samples taken for teduglutide pharmacokinetic (PK) analysis at predose and at 15, 30 minutes and 1, 2, 3, 4, 6, 8, 10, and 12 hours post dose at the first visit that they enter in this study. Subjects enrolling from SHP633-306 will have blood samples taken for teduglutide PK analysis at predose and 1 and 2 hours post dose at the first clinic visit in this study.


06 Nov 2020



In clinic day

Teduglutide

Phone Call

Subjects from SHP633-306: Between V1-V25 study visits occur monthly alternating between clinic visits and phone calls. Starting at V25 clinic visits occur every 3 months. Interim safety visits after PN/IV adjustments are not shown.

Subjects from TED-C14-004: End of study assessments for TED-C14-004 are combined with the SHP633-307 assessments at V1. The study physician will administer the first dose. The study physician must observe the subject administering the study drug in compliance with the study drug administration checklist at least twice before the parent/guardian is allowed to administer the drug without direct observation by the physician. Refer to the criteria for self-administration in the Site Training Guide.

#### **Inclusion and Exclusion Criteria:**

#### **Inclusion Criteria**

Subjects who meet all of the following criterio will be enrolled in this study:

- 1. Ability to voluntarily provide written, signed, and informed consent to participate in the study.
- 2. Completion of the SHP633-306 study or participation in TED-C14-004 Stage 3 or Stage 4.
- 3. Females of childbearing potential must agree to comply with the contraceptive requirements of the protocol.
- 4. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

## **Exclusion Criteria**

There are no exclusion criteria for this study.

## Maximum Duration of Subject Involvement in the Study:

The study will continue until teduglutide is commercially available, the subject's participation in this study is discontinued, or the study is discontinued. The subject's maximum duration of participation is expected to be approximately 3 years. A subject will be considered as having completed the study if the subject has not withdrawn early from the study for any reason prior to completing the end of study (EOS) visit.


**Teduglutide** 06 Nov 2020

#### **Endpoints:**

#### **Efficacy**

The following efficacy endpoints will be assessed at each visit relative to the baseline visit of the relevant core study (SHP633-306 or TED-C14-004):

- Reduction in PN/IV volume of at least 20%
- Absolute and relative change in PN/IV volume
- Complete weaning off PN/IV
- Change in days per week of PN/IV
- Change in plasma citrulline

#### **Pharmacokinetics**

The following parameters will be derived as appropriate (for subjects with rich PK sample collection): area under the plasma concentration-time curve from zero to the last measurable concentration (AUC<sub>0-t</sub>); maximum plasma concentration ( $C_{max}$ ); time to  $C_{max}$  ( $t_{max}$ ); terminal-phase half-life ( $t_{1/2}$ ); apparent clearance (CL/P); and apparent volume of distribution (V/F).

#### Safety

Adverse events (AEs), 12-lead electrocardiogram (ECG), vital signs, laboratory safety data, antibodies to teduglutide, and changes in 48 hour urine output, body weight and body mass index (BMI) will be evaluated. Colonoscopy/sigmoidoscopy will be repeated at Month 24/early termination (ET) and EOS/ET.

#### **Statistical Methods:**

#### **Efficacy**

Efficacy endpoints will be analyzed at each study visit and at the end of study [EOS]), relative to the baseline of the core studies (SHP633-306 and TED-C14-004).

The absolute and percent change in weekly PN/IV volume, days per week of PN/IV support, and plasma citrulline from baseline to each scheduled visit, as well as at EOS, will be summarized using descriptive statistics. The number and percentage of subjects who demonstrate reduction in PN/IV volume of 20% will also be summarized.

The number and percentage of subjects who completely wean off PN/IV support by EOS will be summarized. A subject will be considered to have achieved from PN/IV (completely weaned off PN/IV) if the investigator prescribes no PN/IV at EOS and there is no use of PN/IV recorded in the subject diary during the 2 weeks prior to the last dosing visit.

#### **Pharmacokinetics**

Teduglutide plasma concentrations will be summarized using descriptive statistics (number, mean, standard deviation, minimum, median, and maximum) at nominal time points. Pharmacokinetic parameters will be estimated using non-compartmental analysis as appropriate and summarized using descriptive statistics (number, mean, standard deviation, geometric mean, and CV%, minimum, median, and maximum).

#### Safety

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Treatment-emergent AEs are defined as AEs that started or worsened on or after the date and time of the first dose of study dose. Treatment-emergent AEs will be summarized by system organ class and preferred term using descriptive statistics (eg. number and percentage of subjects). Adverse events will be summarized by severity, relationship to treatment, and for AEs of special interest, AEs leading to discontinuation, and AEs leading to death. Serious AEs will also be tabulated by overall and treatment-related events.

For laboratory tests, 48-hour urine output, vital signs, body weight, BMI, ECG variables, and descriptive statistics (eg, n, mean, standard deviation, median, minimum and maximum values, the number and percentage of subjects in specified categories) will be used to summarize the absolute values and change from baseline at each time point.

The number and percentage of subjects classified as having antibodies to teduglutide will be used to summarize the presence of antibodies.


06 Nov 2020

# STUDY SCHEDULES

Table 1 Schedule of Evaluations and Procedures for Subjects Enrolling from SHP633-306

| | | | | | | | | | | | | 111 | , | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | First<br>Visit <sup>a</sup> | Mo<br>1/13 <sup>b</sup> | Mo<br>2/14 | Mo<br>3/15 <sup>b</sup> | Mo<br>4/16 | Mo<br>5/17 <sup>b</sup> | Mo<br>6/18 | Mo<br>7/19 <sup>b</sup> | Mo<br>8/20 | Mo<br>9/21 <sup>b</sup> | Mo<br>10/22 | Mo<br>11/23 <sup>b</sup> | Mo<br>12 | Mo<br>24 | Every<br>3-Month<br>Visit <sup>c</sup> | EOS/<br>ET |
| Visit Number: | V1 | V2/<br>14 | V3/<br>15 | V4/<br>16 | V5/<br>17 | V6/<br>18 | V7/<br>19 | V8/<br>20 | V9/<br>21 | V10/<br>22 | V11/<br>23 | V12/<br>24 | V13 | V25 | V26 <sup>d</sup> ,<br>V27, etc | EOS/<br>ET |
| Visit Window<br>(days) | | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | .#7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | |
| Informed consent | X | | | | | | | | S | 10) | | | | | | |
| Eligibility | X | | | | | | | | 9 | | | | | | | |
| Medical<br>history <sup>e</sup> | X | | | | | | | 17 5 | | | | | | | | |
| Adverse events | X | X | X | X | X | X | X | X, | X | X | X | X | X | X | X | X |
| Urine pregnancy <sup>f</sup> | X | | X | | X | | χO | ) | X | | X | | X | X | X | X |
| Physical examination <sup>g</sup> | X | | X | | X | : 2 | X | | X | | X | | X | X | X | X |
| Vital signs | X | | X | | X | S.O. | X | | X | | X | | X | X | X | X |
| Body weight | X | | X | | X | 70 | X | | X | | X | | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | |
| Concomitant medications | X | X | X | X | OX. | X | X | X | X | X | X | X | X | X | X | X |
| Safety<br>laboratory tests | X | | X | 40, | X | | X | | X | | X | | X | X | X | X |
| 12-lead ECG | $X^h$ | | 0.0 | | | | X | | | | | | X | X | | X |
| EGD <sup>i</sup> | X | | | | | | | | | | | | | X | | X |
| Colonoscopy/<br>sigmoidoscopy | $X^{j}$ | reg | 0 | | | | | | | | | | | X | | X |
| Citrulline | X 🗸 | 0, | | | | | X | | | | | | X | X | (X) | X |

Table 1 Schedule of Evaluations and Procedures for Subjects Enrolling from SHP633-306

| | | | | | | | | | | | | | 10 | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | First<br>Visit <sup>a</sup> | Mo<br>1/13 <sup>b</sup> | Mo<br>2/14 | Mo<br>3/15 <sup>b</sup> | Mo<br>4/16 | Mo<br>5/17 <sup>b</sup> | Mo<br>6/18 | Mo<br>7/19 <sup>b</sup> | Mo<br>8/20 | Mo<br>9/21 <sup>b</sup> | Mo<br>10/22 | Mo<br>11/23 <sup>b</sup> | Mo<br>12 | Mo<br>24 | Every<br>3-Month<br>Visit <sup>c</sup> | EOS/<br>ET |
| Visit Number: | V1 | V2/<br>14 | V3/<br>15 | V4/<br>16 | V5/<br>17 | V6/<br>18 | V7/<br>19 | V8/<br>20 | V9/<br>21 | V10/<br>22 | V11/<br>23 | V12/<br>24 | V13 | V25 | V26 <sup>d</sup> ,<br>V27, etc | EOS/<br>ET |
| Visit Window<br>(days) | | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ±7 | ±7 | ± 7 | ± 7 | ± 7 | ± 7 | |
| Antibodies to teduglutide <sup>k</sup> | X | | | | | | X | | | . co | | | X | X | (X) | X |
| PK sampling | X <sup>l</sup> | | | | | | | | | | | | | | | |
| Drug<br>dispensing | X | | X | | X | | X | | XS | <b>)</b> , | X | | X | X | X | |
| Interim safety visit <sup>m</sup> | [X] | [X] | [X] | [X] | [X] | [X] | [X] | [X] ? | [X] | [X] | [X] | [X] | [X] | [X] | [X] | [X] |
| Dispense Diary <sup>n</sup> | X | | X | | X | | X | 413 | X | | X | | X | X | X | |
| Review Diary <sup>o</sup> | X | [X] | X | [X] | X | [X] | X | $\mathcal{O}[X]$ | X | [X] | X | [X] | X | X | X | X |
| Record PN/IV<br>use and adjust<br>prescription as<br>indicated | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Teduglutide dosing | $X^p$ | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Confirm<br>administration<br>proficiency | X | | | | COLL | | X | | | | | | X | X | X | |
| Compliance <sup>q</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

(X)=assessment to be performed only every other visit (every 6 months); [X] = Possible interim safety evaluation time point; 48-hour I/O=48-hour fluid intake/urine output; BMI=body mass index; ECG=electrocardiogram; EGD=esophagogastroduodenoscopy; EOS=end of study; EOT=end of treatment; ET=early termination; L=liter; Mo=month; PK=pharmacokinectic; PN/IV=parenteral nutrition/intravenous; V=visit

Note: Clinic visits will alternate with phone visits on a monthly basis for the first 24 months of the extension study for subjects enrolling from SHP633-306.

<sup>&</sup>lt;sup>a</sup> The last visit for SHP633-306 is combined with the first visit for SHP633-307.

<sup>&</sup>lt;sup>b</sup> Subject does not need to visit the clinic. Assessments can be completed over the telephone.

<sup>&</sup>lt;sup>c</sup> Subjects will undergo a chaic visit every 3 months until teduglutide is commercially available, the subject's participation in this study is discontinued, or the study is discontinued.

Table 1 Schedule of Evaluations and Procedures for Subjects Enrolling from SHP633-306

| | | | | | | | | | | | | | 70, | | Every | EOS/ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | First | Mo | Mo | Mo | Mo | Mo | Mo | Mo | Mo | Mo | Mo | Mo | Mo | Mo | 3-Month | ET |
| Procedures | Visit <sup>a</sup> | 1/13 <sup>b</sup> | 2/14 | $3/15^{b}$ | 4/16 | 5/17 <sup>b</sup> | 6/18 | 7/19 <sup>b</sup> | 8/20 | 9/21 <sup>b</sup> | 10/22 | 11/23 <sup>b</sup> | 12 | 24 | Visit <sup>c</sup> | |
| | | V2/ | V3/ | V4/ | V5/ | V6/ | V7/ | V8/ | V9/ | V10/ | V11/ | V12/ | | | V26 <sup>d</sup> , | EOS/ |
| Visit Number: | V1 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 | V13 | V25 | V27, etc | ET |
| Visit Window | | | | | | | | | | | 11/10 | | | | | |
| (days) | | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | ±7 | ± 7 | ± 7 | ± 7 | ± 7 | ± 7 | |

<sup>&</sup>lt;sup>d</sup> Visit 26 will occur 3 months after Visit 25.

<sup>&</sup>lt;sup>e</sup> Updates to the medical history will be collected, consisting of adverse events that were ongoing at the time of completion of SHP633-306, and events that occurred during the period between completion of SHP633-306 and informed consent to SHP 633-307.

<sup>&</sup>lt;sup>f</sup>For women of childbearing potential.

g Full physical examination to be performed at V1, V12, V24, and annually thereafter (V28, V32, V36, etc), and at the EOS/ET visit; a focused examination may be performed at all other clinic visits.

h Electrocardiogram will be conducted for the EOT visit on the previous study (SHP633-306) and if done, the test will not need to be repeated. If the ECG was not conducted for SHP633-306 EOT then the ECG must be conducted within +7 days of the Visit 1 date.

in subjects with risk factors for gastric cancer, EGD is performed at the first clinic visit (VI), Month 24 (V25), and EOS/ET (see Section 7.2.2.6). If the EGD was not conducted for SHP633-306 EOT then the EGD must be conducted within +7 days of the Visit 1 date.

<sup>&</sup>lt;sup>j</sup>Colonoscopy/sigmoidoscopy will be conducted for the EOT visit on the previous study (SHP633-306) and if done, the test will not need to be repeated. If the colonoscopy/sigmoidoscopy was not conducted for SHP633-306 EOT then the colonoscopy/sigmoidoscopy must be conducted within +7 days of the Visit 1 date.

<sup>&</sup>lt;sup>k</sup> Sample for antibody testing must be drawn at least 14 hours after dosing.

<sup>&</sup>lt;sup>1</sup> Subjects enrolling from SHP633-306 will have blood samples taken for PK analysis at predose and 1 and 2 hours post dose at the first clinic visit (V1). If a subject is unable to provide blood samples for PK at the first clinic visit (Visit 1), PK samples can be collected up to 5 days after Visit 1.

m Interim safety evaluations will be performed 5 to 7 days after any change to the subject's PN/IV volume is implemented. Hemoglobin, hematocrit, serum blood urea nitrogen, creatinine, and urine sodium will be measured.

<sup>&</sup>lt;sup>n</sup> The diary is to be completed for the 2-week period prior to every clinic or telephone visit.

<sup>&</sup>lt;sup>o</sup> All subjects will measure 48-hour oral fluid intake and urine output at home immediately prior to the each scheduled visit and interim safety visit. Diary data from the core study may be used for the subject's assessments when entering the SHP633-307 study.

<sup>&</sup>lt;sup>p</sup> The dose of study drug administered at time of entry may be adjusted based on change in the subject's weight from baseline of SHP633-306.

<sup>&</sup>lt;sup>q</sup> Compliance will be checked at every visit by asking subjects if they have taken their study drug according to instructions and by performing drug accountability. Note: The next scheduled visit should be based on the previous visit, not on Visit 1.

Table 2 Schedule of Evaluations and Procedures – For Subjects Enrolling from TED-C14-004

| Procedures | First Visit <sup>a</sup> | Every 3-Month Visit <sup>b</sup> | EOS/ET |
|---|---|---|---|
| Visit Number: | V1 | V1, V2, etc | EOS/ET |
| Visit Window (days) | | ± 7 | ±7 |
| Informed consent | X | | |
| Eligibility | X | | |
| Medical history <sup>c</sup> | X | | 10 |
| Adverse events | X | X | X |
| Urine pregnancy test <sup>d</sup> | X | X | ίζΟΧ |
| Physical examination <sup>e</sup> | X | X | X |
| Vital signs | X | X | X |
| Body weight | X | X | ⊘ X |
| Height | X | 1 | |
| Concomitant medications | X | X XO | X |
| Safety laboratory tests | X | X | X |
| 12-lead ECG | $X^{f}$ | :0 | X |
| EGD <sup>g</sup> | X | | X |
| Colonoscopy/sigmoidoscopy | $X^h$ | 72 | X |
| Citrulline | X | (X) | X |
| Antibodies to teduglutide <sup>i</sup> | X | (X) | X |
| PK sampling | $X^{j}$ | 7 | |
| Drug dispensing | X | X | |
| Interim safety visit k | [X] | [X] | [X] |
| Dispense diary <sup>1</sup> | X | X | |
| Review Diary <sup>m</sup> | X | X | X |
| Record PN/IV use and adjust | X | X | X |
| prescription as indicated | (O) | | |
| Teduglutide dosing | $X^n$ | X | |
| Confirm administration | X <sup>o</sup> X <sup>o</sup> X <sup>o</sup> | (X) | |
| proficiency | | | |
| Compliance <sup>p</sup> | X | X | X |

Property of Lakeda. For I

Table 2 Schedule of Evaluations and Procedures – For Subjects Enrolling from TED-C14-004

| TED-C14-004 | uations and Proced | iures – For Subjects Enr | olling from | 150 |
|---|---|---|---|---|
| Procedures | First Visit <sup>a</sup> | Every 3-Month Visit <sup>b</sup> | EOS/ET | |
| Visit Number: | V1 | V1, V2, etc | EOS/ET | 60. |
| Visit Window (days) | | ± 7 | ± 7 | .03 |

(X)=assessment to be performed only every other visit (every 6 months); [X]=possible interim safety evaluation time point; BMI=body mass index; ECG=electrocardiogram; EGD=esophagogastroduodenoscopy; EOS=end of study; EOT=end of treatment; ET=early termination; L=liter; PK=pharmacokinetic; PN/IV=parenteral nutrition/intravenous; T=time Note: Study visits will be scheduled every 3 months throughout SHP633-307.

Note: The next scheduled visit should be based on the previous visit, not on Visit 1.

<sup>&</sup>lt;sup>a</sup> Assessments for the last visit for TED-C14-004 are combined with the assessments for first visit in SHP633-307, but labs for TED-C14-004 EOS and SHP633-307 V1 need to be drawn for each study.

<sup>&</sup>lt;sup>b</sup> Subjects will undergo a clinic visit every 3 months until teduglutide is commercially available, the subject's participation in this study is discontinued, or the study is discontinued.

<sup>&</sup>lt;sup>c</sup> Updates to the medical history will be collected, consisting of adverse events that were ongoing at the time of completion of TED-C14-004, and events that occurred during the period between completion of TED-C14-004 and informed consent to SHP 633-307.

<sup>&</sup>lt;sup>d</sup> For women of childbearing potential.

e Full physical examination to be performed at V1 and annually thereafter (V5, V9, V13, etc.), and at EOS (or ET) visit; a focused physical examination will be performed at all other study visits.

Electrocardiogram will be conducted for the EOT visit on the previous study (TED-Q14-004) and if done, the test will not need to be repeated. If the ECG was not conducted for TED-C14-004 EOT then the ECG must be conducted within +7 days of the Visit 1 date.

<sup>&</sup>lt;sup>g</sup> Esophagogastroduodenoscopy should be completed at Visit 1 (or conducted within +7 days of the Visit 1 date) for all subjects entering from TED-C14-004. Esophagogastroduodenoscopy is required at EOS/ET for subjects with risk factors for gastric cancer (see Section 7.2.2.6).

h Colonoscopy/sigmoidoscopy will be conducted for the EOT visit on the previous study (TED-C14-004) and if done, the test will not need to be repeated. If the colonoscopy/sigmoidoscopy was not conducted for TED-C14-004 EOT then the colonoscopy/sigmoidoscopy must be conducted within +7 days of the Visit 1 date.

<sup>&</sup>lt;sup>1</sup>Sample for antibody testing must be drawn at least 14 hours after dosing.

<sup>&</sup>lt;sup>j</sup> Subjects enrolling from TED-C14-004 will have blood samples taken for teduglutide PK analysis at predose and at 15, 30 minutes and 1, 2, 3, 4, 6, 8, 10, and 12 hours post dose at the first visit in this study. If a subject is unable to provide blood samples for PK at the first clinic visit (Visit 1), PK samples can be collected up to 5 days after Visit 1.

k Interim safety evaluations will be performed 5 to 7 days after a change to PN/IV volume is implemented. Hemoglobin/hematocrit, serum blood urea nitrogen and serum creatinine, and urine sodium will be measured.

<sup>&</sup>lt;sup>1</sup> The diary is to be completed for the 2-week period prior to every clinic or telephone visit.

m All subjects will measure 48-hour oral fluid intake and urine output at home immediately prior to the next scheduled visit and interim safety visit. Diary data from the core study may be used for the subject's assessments when entering the SHP633-307

<sup>&</sup>lt;sup>n</sup> The dose of study drug administered at time of entry may be adjusted based on change in the subject's weight from baseline of TED-C14-004.

<sup>&</sup>lt;sup>o</sup> The study physician must observe the subject administering the study drug in compliance with the study drug administration checklist at least twice before the subject is allowed to administer the drug without direct observation by the physician. Refer to the criteria for self-administration in the Site Training Guide.

P Compliance will be checked at every visit by asking subjects if they have taken their study drug according to instructions and by performing drug accountability.

#### 1 BACKGROUND INFORMATION

## 1.1 Indication and Current Treatment Options

Short bowel syndrome (SBS) is a rare, serious, disabling, socially incapacitating and potentially life-threatening condition which is the leading cause of intestinal failure (Nightingale and Woodward 2006; Pironi et al. 2015). Intestinal failure from SBS results from surgical resection or congenital defects and is defined as the reduction of gut function below the minimum necessary for the absorption of macronutrients and/or water and electrolytes, such that intravenous supplementation is required to maintain health and/or growth. Patients with SBS are highly prone to malnutrition, diarrhea, dehydration, and an inability to maintain weight due to the reduced intestinal capacity to absorb macronutrients, water, and electrolytes (Dudrick et al. 1991; Nightingale 1999; Rombeau and Rolandelli 1987; Shanbhogue and Molenaar 1994; Vanderhoof and Langnas 1997; Wilmore et al. 1997). Additional potential consequences of SBS include dehydration, electrolyte disturbances, malabsorption of nutrients, gastric hypersecretion, metabolic acidosis, cholelithiasis, nephrolithiasis, steatorrhea, diarrhea, small bowel bacterial overgrowth and weight loss (Nightingale and Woodward 2006; O'keefe et al. 2006).

Following resection, intestinal adaptation may occur in adults during the first 1 to 2 years postsurgery. The adaptive response characterized by mucosal hyperplasia, increased mucosal blood flow, improved segmental absorption and increased hepatobiliary secretions (O'keefe et al. 2006). These morphologic and functional changes are coordinated by the release of glucagon-like peptide 2 (GLP-2) from L-type enteroendocrine cells. In response to lumenal nutrients reaching the distal ileum and colon, L-cells secrete GLP-2, which regulates gastrointestinal secretions, motility, and the local production of additional hormones, cytokines, and growth factors.

The clinical care of SBS is mainly supportive and focuses on optimizing remnant intestinal function through dietary interventions, oral rehydration solutions, antidiarrheal and antisecretory agents. Despite intestinal adaptation following resection, many SBS develop intestinal failure, characterized by the requirement for chronic use of parenteral nutrition/intravenous (PN/IV) or other intravenous fluids to maintain hydration, electrolyte balance, and/or nutritional needs.

Although PN/IV can meet basic nutrition and fluid requirements, it does not improve the body's ability to absorb nutrients. Parenteral nutrition/intravenous dependence is associated with shortened life span (Messing et al. 1999; Scolapio et al. 1999), life threatening complications (eg, sepsis, blood clots, or liver damage), as well as reduced quality of life (Delegge et al. 2007; Jackson and Buchman 2005; Jeppesen 2006). The development of parenteral nutrition-associated liver disease (PNALD) predisposes patients to sepsis, increased mortality rates, and the potential to develop irreversible liver damage (Tazuke and Teitelbaum 2009). The American Gastroenterological Association Medical Position Statement on Short Bowel Syndrome recommends that management of PNALD should include reduction of toxic PN/IV constituents such as phytosterols, a component of soy-based lipid emulsions (American Gastroenterological Association 2003).

The severity of SBS is illustrated by the shortened life-span in patients with moderate to severe disease (Messing et al. 1999). In SBS, survival can be impacted by the underlying condition, by

severe clinical manifestations of malabsorption, and treatment-associated life-threatening complications (O'keefe et al. 2006). With current medical management practices, the overall

In addition, the symptoms of SBS and the inconveniences and complications in relation to PN/IV support may cause potential restrictions in the lifestyle of these patients leading to significant impairment of their quality of life (Jeppesen et al. 1999; Baxter et al. 2014). The impact of SBS and PN/IV on average moving in the lifestyle of the sequence of the sequen average, moving their bowels at least 10 times a day, with multiple ostomy bag changes per day, and having a typical output of 2 to 3 liters of watery diarrhea per day. Patients may be on PN/IV 10 to 15 hours a day for up to 7 days a week. Sleep is disrupted and patients typically cannot work.

#### **Product Background and Clinical Information** 1.2

Teduglutide is a novel, recombinant analog of naturally occurring human GLP-2 that regulates the functional and structural integrity of the cells lining the gastrointestinal (GI) tract. Teduglutide is a 33-amino acid peptide that differs from native GLP-2 in the substitution of glycine for alanine at the second position at the N terminus. As a result, teduglutide demonstrates resistance to degradation by dipeptidyl peptidase 4 and therefore maintains a longer elimination half-life of approximately 2 hours in healthy subjects and 1.3 hours in adult SBS subjects compared to the native peptide, which has a  $t_{1/2}$  of approximately 7 minutes. Teduglutide has been shown in animal studies and previous human clinical trials to increase villus height and crypt depth in the intestinal epithelium, thereby increasing the absorptive surface area of the intestines.

Results of the pivotal study, CL0600-020, showed that teduglutide at a dose of 0.05 mg/kg/day for up to 24 weeks was superior to placebo in reducing PN/IV support in adult subjects with SBS. In this study the responder rate (defined as at least a 20% reduction from baseline in weekly PN/IV volume at Week 20 and Week 24) was 62.8% in the teduglutide 0.05 mg/kg/day group with subjects achieving a mean reduction from baseline in PN/IV volume of 4.4 L/week at Week 24.

In the follow-up long-term extension study CL0600-021, there continued to be evidence of increased efficacy of teduglutide over time in all groups exposed to teduglutide in terms of PN/IV volume reduction, gaining additional days off per week, and achieving complete weaning of parenteral support. The most significant reductions were for those subjects who received 24 weeks of teduglutide 0.05 mg/kg/day in CL0600-020 and continued treatment in CL0600-021 for another 24 months. In this cohort, 10 subjects completely weaned off of PN/IV support and 18/30 (60.0%) had a reduction in their PN/IV requirement of at least 3 days per week. It was encouraging that efficacy was also observed for subjects who initiated treatment in CL0600-021 (ie, those who received placebo or were not treated in CL0600-020).

After only 6 months of treatment, 37.1% of subjects who had received placebo in CL0600-020 had at least a 20% reduction in weekly PN/IV volume, which increased to 55.2% by Month 24.

Two of these subjects completely weaned off of their PN/IV support. In subjects who had not been treated in CL0600-020, 50.0% had at least a 20% reduction in weekly PN/IV volume after 6 months of treatment, which increased to 66.7% by Month 24. One of these subjects completely weaned off of their PN/IV support. Overall, a total of 13 subjects achieved enteral autonomy (independence of PN/IV support), and 25/65 (38.5%) subjects demonstrated a reduction of ≥3 days/week in their parenteral support by the end of study at Month 24. In addition, 21/22 (95.5%) of teduglutide-treated subjects who responded in the previous study maintained their response after an additional 24 months of teduglutide treatment, demonstrating durability of effect. The results of this study support the efficacy of long-term treatment with teduglutide in PN/IV-dependent SBS subjects.

Teduglutide (0.05 mg/kg/day) is currently indicated for the treatment of adult patients with SBS. The European Commission granted a centralized marketing authorization valid throughout the European Union (EU) for teduglutide (REVESTIVE®) on 30 Aug 2012. On 29 Jun 2016, the European Commission granted an extension of the Market Authorization for teduglutide for the ew d and in occumulation of the state of the treatment of patients aged 1 year and above with SBS. A New Drug Application for teduglutide (GATTEX®) was approved by the United States (US) Food and Drug Administration (FDA) on 21 Dec 2012. Teduglutide is currently approved in >30 countries.

#### 2 STUDY OBJECTIVES AND PURPOSE

## 2.1 Rationale for the Study

Teduglutide 0.05 mg/kg/day has demonstrated a favorable benefit-risk profile in clinical studies and is already marketed in the EU and the US. The clinical profile and medical issues related to SBS and PN/IV in Japan are similar to those in the EU and US. Therefore, there is an unmet medical need for Japanese patients with PN/IV-dependent SBS. This study is designed to provide evidence of long-term safety and efficacy of teduglutide in a Japanese SBS patient population.

## 2.2 Study Objectives

ety comple comple complex and subject to the complex of the configuration of the configuration of the configuration of the configuration of the complex complex of the configuration of the configuration of the complex complex of the complex complex of the comple The objectives of this clinical study are to evaluate the long-term safety and efficacy of teduglutide in Japanese subjects with PN/IV-dependent SBS who completed SHP633-306 or

#### 3 STUDY DESIGN

#### 3.1 **Study Design and Flow Chart**

erms of Use This will be a long-term extension study to evaluate the safety and efficacy of teduglutide in Japanese subjects who completed Study SHP633-306 or were in the extension phase of TED-C14-004 (core studies). A schematic representation of the study design is presented in Figure 1.

Once informed consent has been obtained, demographics, updates to medical history and short bowel syndrome history will be obtained. Teduglutide 0.05 mg/kg will be administered once daily until teduglutide is either commercially available, or the subject's participation in this study is discontinued, or the study is discontinued. At each site visit, efficacy (adjustments to PN/IV) and safety will be monitored.

For subjects transitioning from SHP633-306, the SHP633-306 EOS visit assessments will be combined with the assessments for the first visit in SHP633-307. Clinic and phone visits will then alternate on a monthly basis through Month 24; thereafter, clinic visits will occur every 3 months (Table 1). For subjects transitioning from TED-C14-004, the TED-C14-004 EOS visit assessments will be combined with the assessments for the first visit in SHP633-307; thereafter clinic visits will occur every 3 months (Table 2).

Subjects enrolling from TED-C14-004 will have blood samples taken for teduglutide pharmacokinetic (PK) analysis at predose and at 15, 30 minutes and 1, 2, 3, 4, 6, 8, 10, and 12 hours post dose at the first visit that they enter in this study. Subjects enrolling from SHP633-306 will have blood samples taken for teduglutide PK analysis at predose and 1 and 2 hours post dose at the first clinic visit in this study.

#### **Duration and Study Completion Definition** 3.2

The study will continue until teduglutide is commercially available, the subject's participation in this study is discontinued, or the study is discontinued. The subject's maximum duration of participation is expected to be approximately 3 years. A subject will be considered as having completed the study of the subject has not withdrawn early from the study for any reason prior to completing the end of study (EOS) visit.

If teduglutide is approved for marketing, this study will be continued as a post-marketing study. This protocol will continuously be used. "Clinical Study" mentioned in the protocol will be read as "Post-marketing Study" as appropriate.

#### 3.3 **Sites and Regions**

This study is planned to be conducted in approximately 5 sites in Japan.

Figure 1 SHP633-307 Study Schematic



★Self-administration checks

In clinic day

Phone Call

Subjects from SHP633-306: Between V1-V25 study visits occur monthly alternating between clinic visits and phone calls. Starting at V25 clinic visits occur every 3 months. Interim safety visits after PN/IV adjustments are not shown.

Subjects from TED-C14-004: End of study assessments for TED-C14-004 are combined with the SHP633-307 assessments at V1. The study physician will administer the first dose. The study physician must observe the subject administering the study drug in compliance with the study drug administration checklist at least twice before the parent/guardian is allowed to administer the drug without direct observation by the physician. Refer to the criteria for self-administration in the Site Training Guide.

#### 4 STUDY POPULATION

Approximately 5 subjects who completed Study SHP633-306 and up to 7 subjects in TED-C14-004 may enroll in this extension study.

### 4.1 Inclusion Criteria

Subjects who meet all of the following criteria will be enrolled in this study:

- 1. Ability to voluntarily provide written, signed, and informed consent to participate in the study.
- 2. Completion of the SHP633-306 study or participation in TED-C14-004 Stage 3 or Stage 4.
- 3. Females of childbearing potential must agree to comply with the contraceptive requirements of the protocol.
- 4. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

#### 4.2 Exclusion Criteria

There are no exclusion criteria for this study.

## 4.3 Reproductive Potential

To be eligible for treatment with teduglutide, sexually active females of childbearing potential must use a medically acceptable form of contraception. Females of childbearing potential must be advised to use medically acceptable contraceptives throughout the study period and for 30 days following the last dose of investigational product. If hormonal contraceptives are used, they should be administered according to the package insert. Females of childbearing potential who are not currently sexually active must agree to use medically acceptable contraception if they become sexually active during the period of the study and for 30 days following the last dose of investigational product.

Females of childbearing potential must have a negative urine  $\beta$ -HCG pregnancy test at all visits where it is tested to participate in the study (see Section 8.1.6 for information about reporting a pregnancy).

Females of childbearing potential must agree to use medically acceptable methods of contraception at all times during the study and for 30 days following the last dose of investigational product.

## 4.4 Discontinuation of Subjects

A subject may withdraw from the study at any time for any reason without prejudice to their future medical care by the physician or at the institution. The investigator or sponsor may withdraw the subject at any time (eg, in the interest of subject safety). The investigator should

discuss withdrawal of a subject from investigational product with the medical monitor as soon as possible.

If investigational product is discontinued, regardless of the reason, the evaluations listed for EOT/ET are to be performed as completely as possible. Comments (spontaneous or elicited) or complaints pertaining to study drug discontinuation made by the subject must be recorded in the source documents. The reason for termination, date of stopping investigational product, and the total amount of investigational product taken must be recorded in the electronic case report form (eCRF) and source documents. Subjects who discontinue will not be replaced.

#### 4.4.1 **Reasons for Discontinuation**

The reason(s) for permanent discontinuation of treatment and/or withdrawal from the study must be determined by the investigator, and recorded in the subject's medical record and in the eCRF. If a subject is withdrawn for more than 1 reason, each reason should be documented in the source document, and the most clinically relevant reason should be entered in the eCRF.

Reasons for discontinuation include, but are not limited to:

# Protocol deviation Study terminated by sponsor Withdrawal by subject ack of efficacy her S-Subjects "Lost to Follow-up" Prior to Last Scheduled Visit 4.4.2

A minimum of 3 documented attempts must be made to contact any subject lost to follow-up at any time point prior to the last scheduled contact (office visit or telephone contact). At least 1 of these documented attempts must include a written communication sent to the subject's last known address via courier or mail (with an acknowledgement of receipt request) asking that they return to the site for final safety evaluations and return any unused investigational product.

#### 5 CONCOMITANT TREATMENT

#### 5.1 Concomitant Treatment

The administration of all medications including concomitant medications (including prescription and nonprescription medications, dietary and nutritional supplements, and vitamins), study drug, and PN/IV must be recorded from the first visit and for the duration of the study in the appropriate sections of the eCRF. Any diagnostic, surgical or other therapeutic treatments received by a subject during the course of the study will also be recorded on the eCRF. Short term prescriptions lasting less than 72 hours should be recorded in the clinical database as concomitant medications, not as PN/IV adjustments. Examples include fluid resuscitation during treatment of sepsis or acute gastroenteritis, and modification of PN/IV due to interruption of central venous access (PN/IV prescription changes that last 72 hours or more should be recorded in the clinical database as PN/IV adjustments - examples include recurrent replacement of fluid losses, titration of PN/IV due to changes in intestinal absorptive function, and discontinuation of PN/IV due to achievement of enteral autonomy).

The mechanism of action of teduglutide may increase enteral absorption of drugs (eg, motility medication including narcotics and opioids used for the management of SBS, warfarin, psychotropics, metronidazole, digoxin), so consideration should be given to modifying concomitant enteral medication regimens. Titration of concomitant enteral medications should be considered when drugs, especially those with a narrow therapeutic index, are given.

#### **5.1.1** Permitted Treatment

Standard medical therapy for SBS should be continued.

# **5.1.2** Prohibited Treatment

The following medications are prohibited during teduglutide treatment and within the provided timeframe prior to the first visit (Table 3):

**Table 3** Prohibited Treatment

| Prior Therapy | Time Restriction Prior to |
|---|---|
| ۲,0, | the First Visit |
| Glucagon-like peptide-2, human growth hormone, or analogs of these | 6 months |
| Octreotide, dipeptidyl peptidase 4 inhibitors, GLP-1 analogs, and enteral | 30 days |
| glutamine <sup>a</sup> | 30 days |

<sup>&</sup>lt;sup>a</sup> Enteral glutamine refers to L-glutamine powder for oral solution, such as Nutrestore<sup>®</sup> or Endari™, administered in quantities of 5 g or more per dose or more than 10 g per day. The use of elemental formulas that contain glutamine, such as Elental<sup>®</sup>, is allowed.

#### INVESTIGATIONAL PRODUCT 6

containing 5 mg teduglutide as a white lyophilized powder to be reconstituted before use with 0.5 mL sterile water for injection. In addition to the active ingredient (teduglutide), each vial of teduglutide contains L-histidine, mannitol, monobasic sodium phosphate monohydrate. and dibasic sodium phosphate as excipients. Additional information is provided in sterile, single-use 3 mL vials containing 5 mg teduglutide as a white lyophilized powder to be reconstituted before use with 0.5 mL sterile water for injection. In addition to the active ingredient (teduglutide), each vial of teduglutide contains L-histidine, mannitol, monobasic sodium phosphate monohydrate. and dibasic sodium phosphate as excipients. Additional information is provided in sterile, single-use 3 mL vials oly. Shipe application in the ap

#### **Blinding the Treatment Assignment** 6.1.1

Not applicable for this open-label study.

#### **6.2 Administration of Investigational Product**

#### 6.2.1 **Allocation of Subjects to Treatment**

All subjects will receive teduglutide 0.05 mg/kg once daily.

#### 6.2.2 **Dosing**

Teduglutide 0.05 mg/kg once daily will be administered daily by subcutaneous (SC) injection into either thigh or arm or 1 of the 4 quadrants of the abdomen (in subjects without a stoma). Each day, the injection site should be rotated. For subjects with a stoma, the quadrant of the abdomen containing the stoma should not be used. The subject should be dosed at approximately the same time each day. Consecutive doses should be separated by at least 12 hours. The dose of study drug administered at time of entry may be adjusted based on change in the subject's weight from baseline of the core study (SHP633-306 or TED-C14-004). Detailed instructions for reconstitution and injection of the investigational product can be found in the Instructions for Use.

Any subject who achieves complete independence from PN/IV support at any time during the treatment period will continue to receive teduglutide treatment.

#### **Subject Administration** 6.2.2.1

The first dose of teduglutide will be administered by a study physician. The processes for training the subject to self-administer teduglutide and for providing oversight of study drug administration are described in the Site Training Guide. Before a subject is permitted to administer teduglutide, the study physician must observe the subject administering the study drug at least twice in compliance with the teduglutide administration checklist. The checklist is included as an appendix to the Site Training Guide.

After the study physician certifies that the subject can safely administer the study drug, subsequent doses may be administered by the subject at home without direct supervision by the physician. However, at selected study visits during the dosing period (refer to Table 1 for subject enrolling from SHP633-306 and Table 2 for subjects enrolling from TED-C14-004),

administration of the study drug must be performed under direct supervision by the study physician, and the teduglutide administration checklist must be completed again. This ensures that the subject continues to administer the study drug correctly and safely throughout the dosing period.

If at any time a study physician suspects that the subject is no longer capable of administering the study drug safely and accurately, the subject should be reassessed by a study physician using the teduglutide administration checklist. If the subject is deemed unable to administer the study drug, dosing must be performed by a study physician until the subject is retrained and proficiency is confirmed using the teduglutide administration checklist.

Eligibility for teduglutide to be administered by a subject will be judged by a study physician using the following criteria. Refer to the checklist included as an appendix to the Site Training Guide.

Criteria to Initiate Teduglutide Administration by the Subject:

- The subject's condition is stable.
- The subject has been sufficiently trained and is able to administer teduglutide in compliance with the checklist.

Criteria to Discontinue Teduglutide Administration by the Subject:

- The subject is unable to administer teduglutide in compliance with the checklist.
- The subject's condition has deteriorated such that the study physician assesses it is
  inappropriate for the subject to have teduglutide self-administered. In addition to
  discontinuing administration of teduglutide by the subject, if a subject sustains an adverse
  drug reaction where the symptoms are considered intolerable, dose interruption or study
  drug discontinuation should be considered.
- In the study physician's judgment, it is inappropriate for the subject to continue administration of the study drug for any other reason.

## 6.2.3 Unblinding the Treatment Assignment

Not applicable for this open-label study.

# 6.3 Labeling, Packaging, Storage, and Handling

# 6.3.1 Labeling and Packaging

The investigational product will be packaged, labeled, and shipped to the study site by the sponsor or designee. Kits containing 7 vials of investigational product will be provided for this study. The vials will be labeled in accordance with applicable regulatory requirements.

Ancillary kits, containing supplies needed for the reconstitution and administration of the investigational product will also be provided and labeled in accordance with the applicable regulatory requirements.

All investigational product used in this study will be manufactured, tested, labeled, and released according to current legal requirements and Good Manufacturing Practice.

#### 6.3.2 Storage and Handling

The investigator has overall responsibility for ensuring that investigational product is stored in a secure, limited-access location. Limited responsibility may be delegated to the pharmacy or member of the study team, but this delegation must be documented.

Investigational product must be kept in a locked area with access restricted to specific study personnel. Investigational product and ancillary kits will be stored refrigerated at a temperature between 2°C and 8°C (35.6°F to 46.4°F) until dispensed to a subject. The prefilled sterile water for injection syringes will be stored at a temperature between 2°C to 25°C. Once dispensed/supplied to a subject, the investigational product can be stored refrigerated or up to a controlled room temperature (acceptable range of 2°C to 25°C, or 35.6°F to 77°F). The subject will be instructed to keep the investigational product and sterile water diluent at controlled room temperature. If there are concerns that the controlled room temperature cannot be maintained, the investigational product may be refrigerated. The study drug is for single use only, and should be used within 3 hours following reconstitution.

Investigational product must be stored in accordance with labeled storage conditions. Temperature monitoring is required at the storage location to ensure that the investigational product and ancillary kits are maintained within an established temperature range. The investigator is responsible for ensuring that the temperature is monitored throughout the duration of the study and that records are maintained; the temperature should be monitored continuously by using either an in-house system, a mechanical recording device such as a calibrated chart recorder, or by manual means, such that both minimum and maximum thermometric values over a specific time period can be recorded and retrieved as required. Such a device (ie, certified min/max thermometer) would require manual resetting upon each recording. The sponsor must be notified immediately upon discovery of any excursion from the established range. Temperature excursions will require site investigation as to cause and remediation. The sponsor will determine the ultimate impact of excursions on the investigational product and will provide supportive documentation as necessary. Under no circumstances should the product be dispensed to subjects until the impact has been determined and the product is deemed appropriate for use by the sponsor.

The sponsor should be notified immediately if there are any changes to the storage area of the investigational product that could affect the integrity of the product(s), eg, fumigation of a storage room.

Investigational products are distributed by the pharmacy or nominated member of the study team. The pharmacist/nominated team member will enter the unique subject identifier on the investigational product bottle/carton labels, as they are distributed.

## 6.4 Drug Accountability

Investigational product will not be dispatched to the study site until the sponsor or designee has received all required documents from the study site in accordance with applicable regulatory requirements and relevant standard operating procedures. Upon receipt, the study site's pharmacist or delegate is responsible for ensuring that all investigational product received at the site is inventoried and accounted for throughout the study. A copy of the shipping documents must be maintained for the investigator's records. Kits will be shipped to the site once the subject is screened.

Investigators will be provided with sufficient amounts of the investigational product to carry out this protocol for the agreed number of subjects. The investigator or designee will acknowledge receipt of the investigational product, documenting shipment content and condition. Accurate records of all investigational product dispensed, used, returned, and/or destroyed must be maintained as detailed further in this section.

The investigator has overall responsibility for dispensing investigational product. Where permissible, tasks may be delegated to a qualified designee (eg, a pharmacist) who is adequately trained in the protocol and who works under the direct supervision of the investigator. This delegation must be documented in the applicable study delegation of authority form.

The investigator or his/her designee will dispense the investigational product only to subjects included in this study following the procedures set out in the study protocol. Investigational product kits will be dispensed at each of the applicable study visits at which the subject is required to be at the clinic. Each investigational product kit is sufficient for a treatment period of 1 week and enough kits will be supplied to cover the period until the next planned study visit. Additional study kits will be provided as necessary.

Each subject will be given the investigational product according to the protocol. The investigator is to keep a current record of the inventory and dispensing of all clinical supplies. All dispensed medication will be documented on the eCRFs and/or other investigational product record. The investigator is responsible for assuring the retrieval of all study supplies from subjects.

No investigational product stock or returned inventory from a Shire-sponsored study may be removed from the site where originally shipped without prior knowledge and consent by the sponsor. If such transfer is authorized by the sponsor, all applicable local, state, and national laws must be adhered to for the transfer.

The sponsor or its representatives must be permitted access to review the supplies storage and distribution procedures and records.

At the end of the study, or as instructed by the sponsor, all unused stock, subject returned investigational product, and empty/used investigational product packaging are to be sent to the sponsor or designee. The investigator is responsible for assuring the retrieval of all study supplies from subjects.

Returned investigational product must be counted and verified by clinical site personnel and the ible reims of Use sponsor (or study monitor). Shipment return forms, when used, must be signed prior to shipment from the site. Contact the sponsor for authorization to return any investigational product prior to shipment. Shipment of all returned investigational product must comply with local, state, and national laws.

Please see the pharmacy manual for additional information.

#### 6.5 **Subject Compliance**

The subjects must be instructed to bring unused investigational product and empty/used investigational product packaging to every visit. Drug accountability must be assessed and recorded at the container/packaging level for unused investigational product that is contained within the original tamper-evident sealed container (eg, bottles, trays, vials) or at the individual count level for opened containers/packaging.

Subject compliance will be checked by site personnel at every visit by reviewing the subject diaries and asking the subject if he/she has administered the investigational product according to instructions. If any doses have been missed, the reason for missed dose should be documented in the subject's source documentation including, as applicable, the eCRF.

The investigator is responsible for contacting the sponsor or designee when the subject's daily investigational product dosing regimen is interrupted. Attempts should be made to contact the sponsor or designee prior to dose interruption. Reasons for dosage interruption may include but are not limited to hospitalization and adverse events (AEs), a lapse in investigational product delivery, etc.

Subjects who have received 80% of the planned doses administered will be assessed as being Property of Takedai. For non-comm compliant with the study protocol.

#### 7 STUDY PROCEDURES

## 7.1 Study Schedule

Detailed study procedures and assessments to be performed for subjects throughout the study are outlined in the study schedules (Table 1 and Table 2) and must be referred to in conjunction with the instructions provided in this section. The next scheduled visit should be based on the previous visit, not on Visit 1.

Subjects who drop out of the study prior to the final visit should have all early termination procedures done whenever possible.

#### 7.1.1 First Visit

The last visit for SHP633-306/TED-C14-004 may be combined with the first visit for SHP633-307.

Prior to performing any study-related procedures (including those related to Visit 1), the investigator or his/her designee must obtain written informed consent from the subject. The Visit 1 assessments and procedures, beginning with informed consent, will be performed as outlined in Table 1 for subjects transitioning from SHP633-306 and in Table 2 for subjects transitioning from TED-C14-004.

#### 7.1.2 Treatment Period

The treatment period will be performed as outlined in Table 1 and Table 2.

For subjects transitioning from SHP633-306, clinic and phone visits will then alternate on a monthly basis through Month 24; thereafter, clinic visits will occur every 3 months (Table 1). For subjects transitioning from TED-C14-004, clinic visits will occur every 3 months (Table 2).

The study will continue until teduglutide is commercially available, the subject's participation in this study is discontinued, or the study is discontinued.

## 7.2 Study Evaluations and Procedures

## 7.2.1 Efficacy Assessments

# 7.2.1.1 Subject Diaries

Diaries will be provided to subjects. Subjects will record their PN/IV support for 2 weeks prior to each scheduled clinic and interim safety visit. Prior to each scheduled clinic visit and interim safety visit, subjects will also record all enteral fluid intake and urine output over a 48-hour period. Diaries will be distributed to subjects at the time of informed consent and at clinic visits according to the study schedules. Diaries may be completed by the subject or the subject's designee if the subject is physically unable to enter data on his/her own.
## 7.2.1.2 Prescribed Parenteral Nutrition

Adjustments to PN/IV should be based on the guidelines

At the interim visits the PN/IV will be changed if the previous adjustment was not tolerated. Physician-directed changes in a subject's PN/IV volume must be followed by an interim safety visit 5 to 7 days after the adjustment is implemented. If the subject has a AE that prevents him/her from adhering to study requirements, including the PN/IV adjustment algorithm, the subject may be withdrawn from the study.

The prescribed PN/IV weekly total volume and days per week will be recorded. Changes in parenteral support prescription that reflect changes in the subject's intestinal absorption are recorded. Temporary adjustments to parenteral nutrition or IV fluids that last less than 72 hours may be recorded at the discretion of the investigator, but all parenteral support prescriptions that last more than 72 hours must be recorded. The PN/IV constituents are at the discretion of the prescribing physician the identities of parenteral support constituents do not recorded.

## 7.2.1.3 Plasma Citrulline

Plasma citrulline will be measured as an assessment of enterocyte mass. If peripheral venous access is not possible, blood samples for citrulline may be drawn from a central line. The samples will be processed according to instructions in the laboratory manual.

## 7.2.2 Safety Assessments

# 7.2.2.1 Laboratory Evaluations

Safety laboratory tests are to be performed at site visits with results processed by a central laboratory. Although subjects do not need to be in a fasted state at the time of their clinic visit, they should avoid large meals or large volumes of fluid, including PN/IV with lipids, within 3 hours of the clinic visit to permit consistent assessment.

Safety lab tests performed at interim safety visits after PN/IV adjustments will consist of hemoglobin, hematocrit, serum blood urea nitrogen, creatinine, and urine sodium, and may be performed at the investigational site laboratory.

The investigator should assess out-of-range clinical laboratory values for clinical significance, indicating if the value(s) is/are not clinically significant or clinically significant. Abnormal clinical laboratory values, which are unexpected or not explained by the subject's clinical condition, may, at the discretion of the investigator or sponsor, be repeated as soon as possible until confirmed, explained, or resolved. New clinically significant lab tests results should be reported as AEs (see Section 8).

Tests include the following (Table 4):


ermsofuse

06 Nov 2020

# **Table 4** List of Laboratory Tests

## Hematology:

- Hematocrit
- Hemoglobin
- Platelet count
- Red blood cell count
- Red blood cell morphology, if needed
- White blood cell count with differential

## **Urinalysis:**

- Blood
- Glucose
- Leucocytes
- Microscopic analysis
- pH
- Protein
- Specific gravity
- Urine Sodium

# **Pregnancy tests** (females of childbearing potential):

• Urine β-HCG

# **Biochemistry:**

- Albumin
- Alkaline phosphatase
- Alanine aminotransferase
- Amylase
- Aspartate aminotransferase
- Bilirubin (total, direct, and indirect)
- Blood urea nitrogen
- Calcium (total)
- Chloride
- Cholesterol
- Citrulline (plasma)
- C-reactive protein
- Creatinine
- Creatinine clearance
- Gamma-glutamyl transferase
- Glucose
- Lipase
- Magnesium
- Phosphorus
- Potassium
- Sodium
- Triglycerides
- Uric acid

# 7.2.2.2 Antibodies to Teduglutide

Blood samples for analyses of antibodies to teduglutide will be collected. Samples must be drawn at least 14 hours after dosing.

Anti-teduglutide antibody testing is a 3-step process. If a sample tests negative, no further testing is done. If a sample tests positive, further testing is done for teduglutide-specific antibodies. If teduglutide-specific antibodies are detected, the test is deemed "positive" and the titer derived, and neutralizing antibody testing is done. Subjects who test positive for teduglutide-specific antibodies may remain on treatment and blood samples for antibody testing will continue to be collected as per protocol schedule (Table 1 and Table 2).

Blood samples for anti-teduglutide antibody testing may be stored and then analyzed together periodically to streamline the testing procedure. However, if an investigator suspects that a subject is experiencing an AE that may be associated with the development of anti-drug antibodies, relevant samples will be tested for the presence of anti-drug antibodies upon request.

## 7.2.2.3 Physical Examinations

Physical examinations will be performed according to the study schedules to assess the subject's physical status. New clinically significant abnormalities that are detected or diagnosed after study evaluations have begun (after signing of the informed consent) should be recorded on the appropriate AE page of the eCRF. Full physical examination to be performed at first and last visits and on an annual basis; a focused examination will be performed at all other study visits.

# 7.2.2.4 Vital Signs, Body Weight, and Height

Vital signs will be measured according to the study schedules. Measurements will include systolic and diastolic blood pressure (mmHg), pulse rate, body temperature (°C), and height at first visit for all subjects. Blood pressure should be determined by cuff (using the same method, the same arm, and in the same position throughout the study). Subjects should be weighed on the same scale at each study visit. New clinically significant vital sign abnormalities should be recorded on the appropriate AE page of the eCRF.

# 7.2.2.5 Electrocardiograms

A 12-lead ECG will be performed at the study center after the subject has been resting for at least 5 minutes. Results will include general findings only (normal, abnormal-not clinically significant, abnormal-clinically significant). If abnormal, the nature of the abnormality will be collected. Investigators are responsible for providing their own interpretation of the ECG and this will be captured on the eCRF.

Electrocardiogram tracings should be printed signed, and dated by the investigator, and kept with the subject's source documents.

# 7.2.2.6 Gastrointestinal-specific Testing

# COLONOSCOPY/SIGMOIDOSCOPY

For subjects who enter the study from SHP633-306, a colonoscopy/sigmoidoscopy of the remnant colon with polyp removal will be conducted at Visit 1, Visit 25 and EOS/ET. For subjects who enter the study from TED-C14-004, colonoscopy/sigmoidoscopy will be performed at V1 and at EOS/ET. The date and result of colonoscopy are to be recorded in the eCRF.

## **ESOPHAGOGASTRODUODENOSCOPY**

For subjects who enter the study from TED-C14-004, EGD is required at the first clinic visit of SHP633-307. For these subjects, EGD is also required at EOS/ET for subject who present any of the gastric cancer risk factors listed below.

For subjects who enter from SHP633-306, EGD is required at V1,V25, and EOS/ET for subjects who have any of the gastric cancer risk factors listed below.

The gastric cancer risk factors are listed below:

- Age 40 or over at the time of the clinic visit
- History of H pylori gastritis

- History of atrophic gastritis
- History of intestinal metaplasia or dysplasia in the stomach

The dates and results of all EGDs are to be recorded in the eCRF.

## 7.2.2.7 48-Hour Oral Fluid Intake and Urine Output

Subjects will be provided with urine collection containers (as needed) in order to collect 48-hour urine during the 2 days prior to study visits as required. The center staff will contact the subject at least 48 hours before the scheduled visits to remind the subject to start measuring I/O, and to record these measurements into the diary. At these times of 48-hour measurements, the subject should maintain their usual oral fluid intake. These measurements will also be collected at all interim safety visits.

# 7.2.3 Pharmacokinetic Assessments

Subjects enrolling from SHP633-306 will have blood samples taken for teduglutide PK analysis at the first clinic visit (Visit 1)in this study:

- 0-hour (predose) draw: any time prior to the daily dose, on the day of dosing, but at least 14 hours after the previous dose
- 1 hour postdose: ±10 minutes
- 2 hours postdose: ±10 minutes

Subjects enrolling from TED-C14-004 will have blood samples taken for teduglutide PK analysis at the first visit (Visit 1) that they enter in this study:

- 0-hour (predose) draw: any time prior to the daily dose, on the day of dosing, but at least 14 hours after the previous dose
- 15 minutes postdose: ±5 minutes
- 30 minutes postdose. ±5 minutes
- 1 hour postdose. ±10 minutes
- 2 hours postdose: ±10 minutes
- 3 hours postdose: ±10 minutes
- 4 hours postdose: ±30 minutes
- 6 hours postdose: ±30 minutes
- 8 hours postdose: ±30 minutes
- 10 hours postdose: ±30 minutes
- 12 hours postdose: ±30 minutes

Shire

06 Nov 2020

Blood for PK sampling should be collected via peripheral IV or venipuncture, not from a central line. The site of teduglutide administration prior to PK blood draws (arm, thigh, abdomen) and the person administering teduglutide (subject or physician) must be specified.

If a subject is unable to provide blood samples for PK at the first clinic visit (Visit 1), PK samples can be collected up to 5 days after Visit 1.

# 7.3 Changes to Study Procedures Due to a Pandemic

The following information provides guidance regarding changes to the study procedures that could be implemented for study participants or study sites that are impacted by a pandemic (eg, coronavirus disease 2019 [COVID-19] or other future similar unexpected public health concerns) that require physical distancing that may result in subjects missing their visits. This guidance takes references from the FDA Guidance on Conduct of Clinical Trials of Medical Products during COVID-19 Public Health Emergency Guidance for Industry, Investigators, and Institutional Review Boards, March 2020 and updated on 02 July 2020, the European Medicines Agency (EMA) Guidance on the Management of Clinical Trials During the COVID 19 (Coronavirus) Pandemic, Version 3 (28 April 2020), and the EMA Points to consider on implications of Coronavirus disease (COVID-19) on methodological aspects of ongoing clinical trials, dated 26 June 2020.

Because a pandemic (eg, COVID-19) may peak in different regions at different times and restrictions implemented by local laws and recommendations may vary, any decision on procedural changes should be made on a case-by-case basis by the principal investigator, in consultation with the study team (and the medical team as needed), while maintaining patient safety and confidentiality as the priority.

Procedural changes due to COVID-19 (or other similar pandemic) may include the following:

- Informed Consent Form Procedure: If necessary, informed re-consent from a current study participant may be obtained via electronic informed consent capabilities, or an electronic face-to-face consent interview when these individuals are unable to travel to the site, based on local regulations or requirements.
- Clinic / Telephone Visits: In situations where a clinic visit is not completed due to a COVID-19 (or other similar pandemic) concern, a telephone visit may be conducted as an unscheduled safety assessment on subject well-being. The on-site visit will be recorded as "Not Done" with a free text comment referencing COVID-19 (or similar pandemic) and the telephone visit will be documented in the study records and recorded as an unscheduled visit in the eCRF, with a free text comment indicating "Telephone visit".
- Deviations from protocol-specified procedures, eg, missing visits, missing data, alternative visits, etc. will be recorded as related to a pandemic (eg, COVID-19 or other similar pandemic).
- Secure direct-to-patient delivery of the study drug from the investigational site to subjects may be implemented, as per investigational site and sponsor agreement.

Property of Takeda. For non-commercial use only and subject to the applicable Terms of Use

### ADVERSE AND SERIOUS ADVERSE EVENTS ASSESSMENT 8

pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (International Conference on Harmace)

All AEs are collected from the time the informed consent is signed until the defined follow-up period stated in Section 7.1.2. This includes events occurring during the screening phase of the study, regardless of whether or not investigational product is administered. Where possible, a diagnosis rather than a list of symptoms should be recorded. If a diagnosis has not been made, then each symptom should be listed individually. All AEs should be captured on the appropriate AE pages in the eCRF and in source documents. In addition to untoward AEs, unexpected benefits outside the investigational product indication should also be captured on the AE eCRF.

All AEs must be followed to closure (the subject's health has returned to his/her baseline status or all variables have returned to normal), regardless of whether the subject is still participating in the study. Closure indicates that an outcome is reached, stabilization achieved (the investigator does not expect any further improvement or worsening of the event), or the event is otherwise explained. When appropriate, medical tests and examinations are performed so that resolution of event(s) can be documented.

### 8.1.1 **Severity Categorization**

The severity of AEs must be recorded during the course of the event including the start and stop dates for each change in severity. An event that changes in severity should be captured as a new event. Worsening of pretreatment events, after initiation of investigational product, must be recorded as new AEs (for example, if a subject experiences mild intermittent dyspepsia prior to dosing of investigational product, but the dyspepsia becomes severe and more frequent after first dose of investigational product has been administered, a new AE of severe dyspepsia [with the appropriate date of onset] is recorded on the appropriate eCRF).

The medical assessment of severity is determined by using the following definitions:

A type of AE that is usually transient and may require only minimal treatment or

therapeutic intervention. The event does not generally interfere with usual

activities of daily living.

Moderate: A type of AE that is usually alleviated with specific therapeutic intervention. The

event interferes with usual activities of daily living, causing discomfort but poses

no significant or permanent risk of harm to the research subject.

A type of AE that interrupts usual activities of daily living, or significantly affects

clinical status, or may require intensive therapeutic intervention.

# 8.1.2 Relationship Categorization

A physician/investigator must make the assessment of relationship to investigational product for each AE. The investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If there is no valid reason for suggesting a relationship, then the AE should be classified as "not related". Otherwise, if there is any valid reason, even if undetermined or untested, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the AE, then the AE should be considered "related." The causality assessment must be documented in the source document.

The following additional guidance may be helpful:

| Term | Relationship Definition |
|---|---|
| Related | The temporal relationship between the event and the administration of the investigational product is compelling and/or follows a known or suspected response pattern to that product, and the event cannot be explained by the subject's medical condition, other therapies, or accident. |
| Not Related | The event can be readily explained by other factors such as the subject's underlying medical condition, concomitant therapy, or accident and no plausible temporal or biologic relationship exists between the investigational product and the event. |

Adverse events that are related to investigational product that are not resolved at end-of-treatment (EOT) will be followed until the event resolves or stabilizes, as judged by the investigator.

Laboratory values, vital signs, and clinical findings at the scheduled physical examinations must be reported as AEs if the investigator considers the finding to be a clinically significant change from the baseline.

# 8.1.3 Outcome Categorization

The outcome of AEs must be recorded during the course of the study on the eCRF. Outcomes are as follows:

- Fatal
- Not Recovered/Not Resolved
- Recovered/Resolved
- Recovered/Resolved with Sequelae
- Recovering/Resolving
- Unknown

### 8.1.4 **Symptoms of the Disease under Study**

Kerms of Use Symptoms of the disease under study should not be classed as AEs as long as they are within the normal day-to-day fluctuation or expected progression of the disease and are part of the efficacy data to be collected in the study; however, significant worsening of the symptoms should be recorded as an AE.

## 8.1.5 **Clinical Laboratory and Other Safety Evaluations**

A change in the value of a clinical laboratory or vital sign can represent an AE if the change is clinically relevant or if, during treatment with investigational product, a shift of a parameter is observed from a normal value to an abnormal value, or a further worsening of an already abnormal value. When evaluating such changes, the extent of deviation from the reference range, the duration until return to the reference range, either while continuing treatment or after the EOT with the investigational product, and the range of variation of the respective parameter within its reference range, must be taken into consideration.

If, during the study, there are abnormal clinical laboratory values or vital signs which were not present at the pretreatment value observed closest to the start of treatment with teduglutide, further investigations should be done until the values return to within the reference range or until a plausible explanation (eg. concomitant disease) is established for the abnormal values.

The investigator should decide, based on the above criteria and the clinical condition of the subject, whether a change in a clinical laboratory value or vital sign is clinically significant and therefore may represents an AE.

### 8.1.6 **Pregnancy**

All pregnancies are to be reported from the time informed consent is signed until the defined follow-up period stated in Section 7.1.2.

Any report of pregnancy for any female study participant or female partner of male study participant must be reported within 24 hours to IOVIA Services Japan K.K. using the Shire Investigational and Marketed Products Pregnancy Report Form. In the event a subject becomes pregnant during the study, teduglutide administration must be immediately and permanently discontinued.

Every effort should be made to gather information regarding the pregnancy outcome and condition of the infant using the Shire Investigational and Marketed Products Pregnancy Report Form. It is the responsibility of the investigator to obtain this information within 30 calendar days after the initial notification, and approximately 30 calendar days and 1 year postpartum, and report to IQVIA Services Japan K.K.

Pregnancy complications such as spontaneous abortion/miscarriage or congenital abnormality are considered serious adverse events (SAEs) and must be reported using the Shire Clinical Study Adverse Event Form for Serious Adverse Events and Non-serious AEs as Required by Protocol. Note: An elective abortion is not considered an SAE.

In addition to the above, if the investigator determines that complications of the pregnancy meet serious criteria, it must be reported as an SAE using the Shire Clinical Study Adverse Event Form for SAEs and Non-serious AEs as Required by Protocol as well as the Shire Investigational and Marketed Products Pregnancy Report Form. The test date of the first positive serum/urine β-HCG test or ultrasound result will determine the pregnancy onset date.

## 8.1.7 Abuse, Misuse, Overdose, and Medication Error

Abuse, misuse, overdose, or medication error (as defined below) must be reported to the sponsor using the SAE reporting form whether or not they result in an AE/SAE as described in Section 8.2, but such events are only recorded in the eCRF if they result in an AE. Note: The 24-hour reporting requirement for SAEs does not apply to reports of abuse, misuse, overdose, or medication errors unless these result in an SAE.

The categories below are not mutually exclusive; the event can meet more than 1 category.

- Abuse Persistent or sporadic intentional intake of investigational product when used for a non-medical purpose (eg, to alter one's state of consciousness or get high) in a manner that may be detrimental to the individual and/or society.
- Misuse Intentional use of investigational product other than as directed or indicated at any dose (Note: this includes a situation where the investigational product is not used as directed at the dose prescribed by the protocol).
- Overdose Administration of the investigational product at a dose or frequency greater than 0.05 mg/kg subcutaneous once daily. An overdose occurs if any of the following criteria are met:
  - More than 0.05 mg/kg is given at any one time
  - Consecutive doses are spaced less than 12 hours apart
  - Any more than 0.05 mg/kg in one day (a day is defined as beginning at 12:00 AM and ending at 11:59 PM)
- Medication Error —An error made in prescribing, dispensing, administration, and/or use of an investigational product. For studies, medication errors are reportable to the sponsor only as defined below.
  - Cases of subjects missing doses of the investigational product are not considered reportable as medication errors.
  - Medication errors should be collected/reported for all products under investigation.
  - The administration and/or use of an expired investigational product should be considered as a reportable medication error.

All investigational product provided to pediatric subjects should be supervised by the parent/legally authorized representative/caregiver.

### 8.2 **Serious Adverse Event Procedures**

### 8.2.1 **Reference Safety Information**

The reference for safety information for this study is the investigator's brochure which the sponsor has provided under separate cover to all investigators.

### 8.2.2 **Reporting Procedures**

rems of Use All initial and follow-up SAE reports must be reported by the investigator to the sponsor or designee within 24 hours of the first awareness of the event. Note: The 24-hour reporting requirement for SAEs does not apply to reports of abuse, misuse, overdose, or medication errors (see Section 8.1.7) unless they result in an SAE.

All Adverse Events of Special Interest, as defined in Section 8.3, must be reported by the investigator to the sponsor or designee within 24 hours of the first awareness of the event even if the event does not fulfill seriousness criterion.

The investigator must complete, sign, and date the Shire Clinical Study Adverse Event Form for Serious Adverse Events (SAEs) and Non-serious AEs as Required by Protocol and verify the accuracy of the information recorded on the form with the corresponding source documents (Note: Source documents are not to be sent unless requested). The investigator must fax or e-mail the completed form to IQVIA Services Japan K.K. Applicable fax numbers and email addresses are found in the Emergency Contact Information.

### **Serious Adverse Event Definition** 8.2.3

An SAE is any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose:

- Results in death
- Is life-threatening. Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it was more severe.
- Requires inpatient hospitalization or prolongation of existing hospitalization. Note: Hospitalizations, which are the result of elective or previously scheduled surgery for preexisting conditions, which have not worsened after initiation of treatment, should not be classified as SAEs. For example, an admission for a previously scheduled ventral hernia repair would not be classified as an SAE; however, complication(s) resulting from a hospitalization for an elective or previously scheduled surgery that meet(s) serious criteria must be reported as SAE(s).
- Results in persistent or significant disability/incapacity.
- Is a congenital abnormality/birth defect.
- Is an important medical event. Note: Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or

surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home; blood dyscrasias or convulsions that do not result in inpatient hospitalization; or the development of drug dependency or drug abuse.

### 8.2.4 Serious Adverse Event Collection Time Frame

ns of Use All SAEs (regardless of relationship to study) are collected from the time the informed consent is obtained until the defined follow-up period stated in Section 7.1.2, and must be reported to the sponsor or designee within 24 hours of the first awareness of the event.

In addition, any SAE(s) considered "related" to the investigational product and discovered by the investigator at any interval after the study has completed must be reported to the sponsor or designee within 24 hours of the first awareness of the event.

### 8.2.5 **Serious Adverse Event Onset and Resolution Dates**

The onset date of the SAE is defined as the date the event meets serious criteria. The resolution date is the date the event no longer meets serious criteria, the date the symptoms resolve, or the event is considered chronic. In the case of hospitalizations, the hospital admission and discharge dates are considered the onset and resolution dates, respectively.

In addition, any signs or symptoms experienced by the subject after signing the informed consent form, or leading up to the onset date of the SAE, or following the resolution date of the SAE, must be recorded as an AE, if appropriate.

### 8.2.6 **Fatal Outcome**

Any SAE that results in the subject's death (ie, the SAE was noted as the primary cause of death) must have fatal checked as an outcome with the date of death recorded as the resolution date. For all other events ongoing at the time of death that did not contribute to the subject's death, the outcome should be considered not resolved, without a resolution date recorded.

For any SAE that results in the subject's death or any ongoing events at the time of death, unless another investigational product action was previously taken (eg, drug interrupted, reduced, withdrawn), the action taken with the investigational product should be recorded as "dose not changed" or "not applicable" (if the subject never received investigational product). The investigational product action of "withdrawn" should not be selected solely as a result of the subject's death.

# Regulatory Agency, Institutional Review Board, Ethics Committee, and Site Reporting

The sponsor is responsible for notifying the relevant regulatory authorities of related, unexpected SAEs.

In addition, the sponsor and/or designee is responsible for notifying active sites of all related, unexpected SAEs occurring during all interventional studies across the teduglutide program.

The investigator is responsible for notifying the local Institutional Review Board (IRB) or the relevant local regulatory authority of all SAEs that occur at his or her site as required.

An AE of special interest is an AE (serious or nonserious) of scientific and medical concern specific to the sponsor's product or program and for which ongoing monitoring and immediate notification by the investigator to the sponsor is required.

The AEs of special interest that require expedited regulators:
following:

- Benign neoplasia of the GI tract including the hepatobiliary system

  Tumor-promoting ability (eg, benign and/or malignant neoplasia of those of the GI or hepatobiliary system) Tumor-promoting ability (eg, benign and/or malignant neoplasia of any kind, not limited to

must b .s describe only and and second of takeda. For noncommercial use only and property of takeda. For AEs of special interest, the sponsor or designee must be informed within 24 hours of first awareness as per the SAE notification instructions described in Section 8.2.2 even if the event

## 9 DATA MANAGEMENT AND STATISTICAL METHODS

## 9.1 Data Collection

The investigators' authorized site personnel must enter the information required by the protocol on the eCRF. A study monitor will visit each site in accordance with the monitoring plan and review the eCRF data against the source data for completeness and accuracy. Discrepancies between source data and data entered on the eCRF will be addressed by qualified site personnel. When a data discrepancy warrants correction, the correction will be made by authorized site personnel. Data collection procedures will be discussed with the site at the site initiation visit and/or at the investigator's meeting. Once a subject is enrolled, it is expected that site personnel will complete the eCRF entry within approximately 3 business days of the subject's visit.

## 9.2 Clinical Data Management

Data are to be entered into a clinical database as specified in the data management plan. Quality control and data validation procedures are applied to ensure the validity and accuracy of the clinical database.

Data are to be reviewed and checked for omissions, errors, and values requiring further clarification using computerized and manual procedures. Data queries requiring clarification are to be communicated to the site for resolution. Only authorized personnel will make corrections to the clinical database, and all corrections are documented in an auditable manner.

# 9.3 Statistical Analysis Process

The data collected in this study will be analyzed by the sponsor or designee. All statistical analyses will be performed using SAS® (SAS Institute, Cary, NC, US) version 9.3 or higher.

The statistical analysis plan (SAP) will provide the statistical methods and definitions for the analysis of the efficacy and safety data, as well as describe the approaches to be taken for summarizing other study information such as subject disposition, demographics and baseline characteristics, investigational product exposure, and prior and concomitant medications. The SAP will also include a description of how missing, unused and spurious data will be addressed.

No claims of statistical significance will be made; however, 95% confidence intervals will be provided, if applicable. Continuous variables, including those assessed on a discrete scale, will be summarized using descriptive statistics including number of subjects, mean, median, standard deviation, maximum, and minimum. For categorical variables, statistical summaries will include number of subjects and percentages. The derivations of the weekly PS volume will be described in the study statistical analysis plan in detail.

## 9.4 Planned Interim Analysis

An interim analysis will be conducted when the last subject who enters the study from SHP633-306 reaches the Month 6 visit (Visit 7) and the last subject from TED-C14-004 reaches Visit 1. Additional interim analyses may be conducted during the study, as needed.

Analyses will be descriptive in nature. No formal comparisons are planned and no hypotheses will be formally tested. Due to the open-label nature of this study, personnel involved in

The number of subjects in this study is not based on statistical power considerations as this is an extension study of the core study SHP633-306 and TED-C14-004. Approximately 5 subjects who completed Study SHP633-306 and 7 subjects in the extension about this extension study.

### 9.6 **Study Population**

The safety population will include all enrolled subjects in the study. A subject will be considered enrolled in the study once the informed consent has been obtained and the subject meets all of the study inclusion criteria. Safety population will be used for both safety and efficacy analyses.

The pharmacokinetic population will include all subjects who receive at least 1 dose of teduglutide and have at least 1 evaluable post-dose pharmacokinetic concentration value.

## 9.7 **Efficacy Analyses**

The following efficacy endpoints will be analyzed at each study visit and at the EOS, relative to the baseline of the core studies (SHP633-306 and TED-C14-004):

- Reduction in PN/IV volume of at least 20%
- Absolute and relative change in PN/IV volume
- Complete weaning off PN/IV
- Change in days per week of PN/IV
- Change in plasma citrulline

The absolute and percent change in weekly PN/IV volume, days per week of PN/IV support, and plasma citrulline from baseline to each scheduled visit, as well as at EOS, will be summarized using descriptive statistics. The number and percentage of subjects who demonstrate reduction in PN/IV volume of 20% will also be summarized.

The number and percentage of subjects who completely wean off PN/IV support by EOS will be summarized. A subject will be considered to have achieved from PN/IV (completely weaned off PN/IV) if the investigator prescribes no PN/IV at EOS and there is no use of PN/IV recorded in the subject diary during the 2 weeks prior to the last dosing visit.

# 9.8 Safety Analyses

The safety endpoints include AEs, 12-lead ECG, vital signs, laboratory safety data, antibodies to teduglutide, and 48-hour urine output, body weight, BMI and gastrointestinal-specific tests.

Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Treatment-emergent AEs are defined as AEs that started or worsened on or after the date and time of the first dose of study dose. Treatment-emergent AEs will be summarized by system organ class and preferred term using descriptive statistics (eg, number and percentage of subjects). Adverse events will be summarized by severity, relationship to treatment, and for AEs of special interest, AEs leading to discontinuation, and AEs leading to death. Serious AEs will also be tabulated by overall and treatment-related events.

For laboratory tests, 48-hour urine output, vital signs, body weight, BMI, EGG variables, and descriptive statistics (eg, n, mean, standard deviation, median, minimum and maximum values, the number and percentage of subjects in specified categories) will be used to summarize the absolute values and change from baseline at each time point.

The number and percentage of subjects classified as having antibodies to teduglutide will be used to summarize the presence of antibodies.

# 9.9 Pharmacokinetics Analyses

Teduglutide plasma concentrations will be summarized using pharmacokinetic population with descriptive statistics (number, mean and standard deviation, minimum, median, and maximum) at nominal time points.

The following PK parameters will be derived as appropriate (for subjects with rich PK sample collection): area under the plasma concentration-time curve from zero to the last measurable concentration (AUC<sub>0-t</sub>); maximum plasma concentration (C<sub>max</sub>); time to C<sub>max</sub> (t<sub>max</sub>); terminal-phase half-life (t<sub>1/2</sub>); apparent clearance (CL/F); and apparent volume of distribution (V/F) and summarized using descriptive statistics (number, mean, standard deviation, geometric mean, and CV%, minimum, median, and maximum).

### SPONSOR'S AND INVESTIGATOR'S RESPONSIBILITIES 10

Terms of Use This study is conducted in accordance with current applicable regulations, ICH, EU Directive 2001/20/EC and its updates, and local ethical and legal requirements.

The name and address of each third-party vendor (eg. contract research organization [CRO]) used in this study will be maintained in the investigator's and sponsor's files, as appropriate.

### 10.1 **Sponsor's Responsibilities**

### 10.1.1 **Good Clinical Practice Compliance**

The study sponsor and any third party to whom aspects of the study management or monitoring have been delegated will undertake their assigned roles for this study in compliance with all applicable industry regulations, ICH Good Clinical Practice (GCP) Guideline E6 (1996), EU Directive 2001/20/EC, as well as all applicable national and local laws and regulations.

Visits to sites are conducted by representatives of the study sponsor and/or the company organizing/managing the research on behalf of the sponsor to inspect study data, subjects' medical records, and eCRFs in accordance with current GCP and the respective local and (inter)national government regulations and guidelines. Records and data may additionally be reviewed by auditors or by regulatory authorities.

The sponsor ensures that local regulatory authority requirements are met before the start of the study. The sponsor (or a nominated designee) is responsible for the preparation, submission, and confirmation of receipt of any regulatory authority approvals required prior to release of investigational product for shipment to the site.

### Indemnity/Liability and Insurance 10.1.2

The sponsor of this research adheres to the recommendations of the Association of British Pharmaceutical Industry Guidelines. If appropriate, a copy of the indemnity document is supplied to the investigator before study initiation, per local country guidelines.

The sponsor ensures that suitable clinical study insurance coverage is in place prior to the start of the study. An insurance certificate is supplied, as necessary.

## **Public Posting of Study Information** 10.1.3

The sponsor is responsible for posting appropriate study information on applicable websites. Information included in clinical study registries may include participating investigators' names and contact information.

## 10.1.4 Submission of Summary of Clinical Study Report to Competent Authorities of Member States Concerned and Ethics Committees

The sponsor will provide a summary of the clinical study report to the competent authority of the member state(s) concerned as required by regulatory requirement(s) and to comply with the Community guideline on GCP. This requirement will be fulfilled within 6 months of the end of

the study completion date for pediatric studies and within 1 year for non-pediatric studies as per guidance.

## 10.1.5 Study Suspension, Termination, and Completion

The sponsor may suspend or terminate the study, or part of the study, at any time for any reason. If the study is suspended or terminated, the sponsor will ensure that applicable sites, regulatory agencies and IRBs/ECs are notified as appropriate. Additionally, the discontinuation of a registered clinical study which has been posted to a designated public website will be updated accordingly.

# 10.2 Investigator's Responsibilities

## **10.2.1** Good Clinical Practice Compliance

The investigator must undertake to perform the study in accordance with ICH GCP Guideline E6 (1996), EU Directive 2001/20/EC, and applicable regulatory requirements and guidelines.

It is the investigator's responsibility to ensure that adequate time and appropriately trained resources are available at the site prior to commitment to participate in this study. The investigator should also be able to estimate or demonstrate a potential for recruiting the required number of suitable subjects within the agreed recruitment period.

The investigator will maintain a list of appropriately qualified persons to whom the investigator has delegated significant study-related tasks, and shall, upon request of the sponsor, provide documented evidence of any licenses and certifications necessary to demonstrate such qualification. Curriculum vitae for investigators and sub investigators are provided to the study sponsor (or designee) before starting the study.

If a potential research subject has a primary care physician, the investigator should, with the subject's consent, inform them of the subject's participation in the study.

# 10.2.2 Protocol Adherence and Investigator Agreement

The investigator and any co-investigators must adhere to the protocol as detailed in this document. The investigator is responsible for enrolling only those subjects who have met protocol eligibility criteria. Investigators are required to sign an investigator agreement to confirm acceptance and willingness to comply with the study protocol.

If the investigator suspends or terminates the study at their site, the investigator will promptly inform the sponsor and the IRB/EC and provide them with a detailed written explanation. The investigator will also return all investigational product, containers, and other study materials to the sponsor. Upon study completion, the investigator will provide the sponsor, IRB/EC, and regulatory agency with final reports and summaries as required by (inter)national regulations.

Communication with local IRBs/ECs, to ensure accurate and timely information is provided at all phases during the study, may be done by the sponsor, applicable CRO, investigator, or for multicenter studies, the coordinating principal investigator according to national provisions and will be documented in the investigator agreement.

### 10.2.3 **Documentation and Retention of Records**

### 10.2.3.1 **Electronic Case Report Forms**

Electronic case report forms are supplied by the sponsor or designe and should be handled in accordance with instructions from the sponsor.

KINS OF USE The investigator is responsible for maintaining adequate and accurate medical records from which accurate information is recorded onto eCRFs, which have been designed to record alk observations and other data pertinent to the clinical investigation. Case report forms must be completed by the investigator or designee as stated in the site delegation log. All data will have separate source documentation; no data will be recorded directly onto the eCRF.

All data sent to the sponsor must be endorsed by the investigator. The study monitor will verify the contents against the source data per the monitoring plan. If the data are unclear or contradictory, queries are sent for corrections or verification of data.

## Recording, Access, and Retention of Source Data and Study Documents 10.2.3.2

Original source data to be reviewed during this study will include, but are not limited to: subject's medical file, subject diaries, original clinical laboratory reports, and imaging reports.

All key data must be recorded in the subject's medical records.

The investigator must permit authorized representatives of the sponsor; the respective national, local, or foreign regulatory authorities; the IRB/EC; and auditors to inspect facilities and to have direct access to original source records relevant to this study, regardless of media.

The study monitor (and auditors, IRB/EC or regulatory inspectors) may check the eCRF entries against the source documents. The consent form includes a statement by which the subject agrees to the monitor/auditor from the sponsor or its representatives, national or local regulatory authorities, or the IRB/EC, having access to source data (eg, subject's medical file, appointment books, original laboratory reports, X-rays etc).

These records must be made available within reasonable times for inspection and duplication, if required, by a properly authorized representative of any regulatory agency (eg, the US FDA, EMA, UK Medicines and Healthcare products Regulatory Agency) or an auditor.

Essential documents must be maintained according to ICH GCP requirements and may not be destroyed without written permission from the sponsor.

### 10.2.3.3 Audit/Inspection

To ensure compliance with relevant regulations, data generated by this study must be available for inspection upon request by representatives of, for example, the US FDA (as well as other US national and local regulatory authorities), the EMA, the Medicines and Healthcare products Regulatory Agency, other regulatory authorities, the sponsor or its representatives, and the IRB/EC for each site.

## 10.2.3.4 Financial Disclosure

The investigator is required to disclose any financial arrangement during the study and for 1 year after, whereby the outcome of the study could be influenced by the value of the compensation for conducting the study, or other payments the investigator received from the sponsor. The following information is collected: any significant payments from the sponsor or subsidiaries such as a grant to fund ongoing research, compensation in the form of equipment, retainer for ongoing consultation or honoraria; any proprietary interest in investigational product; any significant equity interest in the sponsor or subsidiaries as defined in 21 CFR 54 2(b) (1998).

## 10.3 Ethical Considerations

## 10.3.1 Informed Consent

It is the responsibility of the investigator to obtain written informed consent from all study subjects prior to any study-related procedures including screening assessments. All consent documentation must be in accordance with applicable regulations and GCP. Each subject or the subject's legally authorized representative, as applicable, is requested to sign and date the subject informed consent form or a certified translation if applicable, after the subject has received and read (or been read) the written subject information and received an explanation of what the study involves, including but not limited to: the objectives, potential benefits and risk, inconveniences, and the subject's rights and responsibilities. A copy of the informed consent documentation (ie, a complete set of subject information sheets and fully executed signature pages) must be given to the subject or the subject's legally authorized representative, as applicable. This document may require translation into the local language. Signed consent forms must remain in each subject's study file and must be available for verification at any time.

The principal investigator provides the sponsor with a copy of the consent form that was reviewed by the IRB/EC and received their favorable opinion/approval. A copy of the IRB/EC's written favorable opinion/approval of these documents must be provided to the sponsor prior to the start of the study unless it is agreed to and documented (abiding by regulatory guidelines and national provisions) prior to study start that another party (ie, sponsor or coordinating principal investigator) is responsible for this action. Additionally, if the IRB/EC requires modification of the sample subject information and consent document provided by the sponsor, the documentation supporting this requirement must be provided to the sponsor.

## 10.3.2 Institutional Review Board or Ethics Committee

For sites outside the EU, it is the responsibility of the investigator to submit this protocol, the informed consent document (approved by the sponsor or their designee), relevant supporting information and all types of subject recruitment information to the IRB/EC for review, and all must be approved prior to site initiation.

The applicant for an EC opinion can be the sponsor or investigator for sites within the EU; for multicenter studies, the applicant can be the coordinating principal investigator or sponsor, according to national provisions.

Responsibility for coordinating with IRBs/ECs is defined in the investigator agreement.

Prior to implementing changes in the study, the sponsor and the IRB/EC must approve any revisions of all informed consent documents and amendments to the protocol unless there is a subject safety issue.

Investigational product supplies will not be released until the sponsor/designee has received written IRB/EC approval of and copies of revised documents.

ins of Use For sites outside the EU, the investigator is responsible for keeping the IRB/EC apprised of the progress of the study and of any changes made to the protocol, but in any case at least once a year; this can be done by the sponsor or investigator for sites within the EU, or for multicenter studies, it can be done by the coordinating principal investigator, according to national provisions. The investigator must also keep the local IRB/EC informed of any serious and significant AEs.

### 10.4 **Privacy and Confidentiality**

The confidentiality of records that may be able to identify subjects will be protected in accordance with applicable laws, regulations, and guidelines.

After subjects have consented to take part in the study, the sponsor and/or its representatives reviews their medical records and data collected during the study. These records and data may, in addition, be reviewed by others including the following: independent auditors who validate the data on behalf of the sponsor; third parties with whom the sponsor may develop, register, or market teduglutide; national or local regulatory authorities; and the IRB(s)/EC(s) which gave approval for the study to proceed.

The sponsor and/or its representatives accessing the records and data will take all reasonable precautions in accordance with applicable laws, regulations, and guidelines to maintain the confidentiality of subjects' identities.

Subjects are assigned a unique identifying number; however, their initials and date of birth may also be collected and used to assist the sponsor to verify the accuracy of the data (eg., to confirm that laboratory results have been assigned to the correct subject).

The results of studies – containing subjects' unique identifying number, relevant medical records, and possibly initials and dates of birth – will be recorded. They may be transferred to, and used in other countries which may not afford the same level of protection that applies within the countries where this study is conducted. The purpose of any such transfer would include: to support regulatory submissions, to conduct new data analyses to publish or present the study results, or to answer questions asked by regulatory or health authorities.

## 10.5 **Study Results/Publication Policy**

Shire will endeavor to publish the results of all qualifying, applicable, and covered studies according to external guidelines in a timely manner regardless of whether the outcomes are perceived as positive, neutral, or negative. Additionally, Shire adheres to external guidelines (eg, Good Publication Practices) when forming a publication steering committee, which is done for

large, multicenter Phase 2 to 4 and certain other studies as determined by Shire. The purpose of the publication steering committee is to act as a non-commercial body that advises or decides on dissemination of scientific study data in accordance with the scope of this policy.

All publications relating to Shire products or projects must undergo appropriate technical and intellectual property review, with Shire agreement to publish prior to release of information. The review is aimed at protecting the sponsor's proprietary information existing either at the commencement of the study or generated during the study. To the extent permitted by the publisher and copyright law, the principal investigator will own (or share with other authors) the copyright on his/her publications. To the extent that the principal investigator has such sole, joint or shared rights, the principal investigator grants the sponsor a perpetual, irrevocable, royalty free license to make and distribute copies of such publications.

The term "publication" refers to any public disclosure including original research articles, review articles, oral presentations, abstracts and posters at medical congresses, journal supplements, letters to the editor, invited lectures, opinion pieces, book chapters, electronic postings on medical/scientific websites, or other disclosure of the study results in printed, electronic, oral or other form.

Subject to the terms of the paragraph below, the investigator shall have the right to publish the study results, and any background information provided by the sponsor that is necessary to include in any publication of study results, or necessary for other scholars to verify such study results. Notwithstanding the foregoing, no publication that incorporates the sponsor's confidential information shall be submitted for publication without the sponsor's prior written agreement to publish and shall be given to the sponsor for review at least 60 days prior to submission for publication.

If requested in writing by Shire, the institution and principal investigator shall withhold submission of such publication for up to an additional 60 days to allow for filing of a patent application.

If the study is part of a multicenter study, the first publication of the study results shall be made by the sponsor in conjunction with the sponsor's presentation of a joint, multicenter publication of the compiled and analyzed study results. If such a multicenter publication is not submitted to a journal for publication by the sponsor within an 18-month period after conclusion, abandonment, or termination of the study at all sites, or after the sponsor confirms there shall be no multicenter study publication of the study results, an investigator may individually publish the study results from the specific site in accordance with this section. The investigator must, however, acknowledge in the publication the limitations of the single site data being presented.

Unless otherwise required by the journal in which the publication appears, or the forum in which it is made, authorship will comply with the International Committee of Medical Journal Editors (ICMJE) current standards. Participation as an investigator does not confer any rights to authorship of publications.

is of Use

**Teduglutide** 

**REFERENCES** 

Shire

11

- American Gastroenterological Association 2003. American Gastroenterological Association medical position statement: short bowel syndrome and intestinal transplantation. Gastroenterology, 124, 1105-1110.
- Amiot, A., Messing, B., Corcos, O., Panis, Y. & Joly, F. 2013. Determinants of home parenteral nutrition dependence and survival of 268 patients with non-malignant short bowel syndrome Clin Nutr, 32, 368-74.
- Baxter, J. P., Fayers, P. M. & Mckinlay, A. W. 2006. A review of the quality of life of adult patients treated with long-term parenteral nutrition. Clin Nutr, 25, 543-53.
- Delegge, M., Alsolaiman, M. M., Barbour, E., Bassas, S., Siddiqi, M. F. & Moore, N. M. 2007. Short bowel syndrome: parenteral nutrition versus intestinal transplantation. Where are we today? Dig Dis Sci, 52, 876-92.
- Dudrick, S. J., Latifi, R. & Fosnocht, D. E. 1991. Management of the short-bowel syndrome. Surg Clin North Am, 71, 625-43.
- Jackson, C. & Buchman, A. L. 2005. Advances in the management of short bowel syndrome. Curr Gastroenterol Rep. 7, 373-8.
- Jeppesen, P. B. 2006. Glucagon-like peptide-2: update of the recent clinical trials. Gastroenterology, 130, S127-31.
- Jeppesen, P. B., Langholz, E. & Mortensen, P. B. 1999. Quality of life in patients receiving home parenteral nutrition. Gut, 44, 844-52.
- Messing, B., Crenn, P., Beau, P., Boutron-Ruault, M. C., Rambaud, J. C. & Matuchansky, C. 1999. Long-term survival and parenteral nutrition dependence in adult patients with the short bowel syndrome. Gastroenterology, 117, 1043-50.
- Nightingale, J. & Woodward, J. M. 2006. Guidelines for management of patients with a short bowel. Gut, 55 Suppl 4, iv1-12.
- Nightingale, J. M. 1999. Management of patients with a short bowel. Nutrition, 15, 633-7.
- O'keefe, S. J., Buchman, A. L., Fishbein, T. M., Jeejeebhoy, K. N., Jeppesen, P. B. & Shaffer, J. 2006. Short bowel syndrome and intestinal failure: consensus definitions and overview. Clin Gastroenterol Hepatol, 4, 6-10.
- Pironi, L., Arends, J., Baxter, J., Bozzetti, F., Pelaez, R. B., Cuerda, C., Forbes, A., Gabe, S., Gillanders, L., Holst, M., Jeppesen, P. B., Joly, F., Kelly, D., Klek, S., Irtun, O., Olde Damink, S. W., Panisic, M., Rasmussen, H. H., Staun, M., Szczepanek, K., Van Gossum, A., Wanten, G., Schneider, S. M. & Shaffer, J. 2015. ESPEN endorsed recommendations. Definition and classification of intestinal failure in adults. Clin Nutr, 34, 171-80.

- Rombeau, J. L. & Rolandelli, R. H. 1987. Enteral and parenteral nutrition in patients with enteric fistulas and short bowel syndrome. Surg Clin North Am, 67, 551-71.
- Shanbhogue, L. K. & Molenaar, J. C. 1994. Short bowel syndrome: metabolic and surgical management. Br J Surg, 81, 486-99.

  Tazuke, Y. & Teitelbaum, D. H. 2009. Alteration of care total parenteral nutrition. I Padi:

- Vanderhoof, J. A. & Langnas, A. N. 1997. Short-bowel syndrome in children and adults. Gastroenterology, 113, 1767-78.
- Wilmore, D. W., Byrne, T. A. & Persinger, R. L. 1997. Short bowel syndrome: New therapeutic approaches. Current Problems in Surgery, 34, 389,391-444.
- Property of Takeda. For noncommercial use only of Takeda. Winkler, M. F. & Smith, C. E. 2014. Clinical, social, and economic impacts of home parenteral nutrition dependence in short bowel syndrome. JPENJ Parenter Enteral Nutr, 38, 32s-37s.





Property of Takeda. For non-commercial use only and subject to the





Property of Lakedai.



Property of Takedai. For I